

« Etude sur l'observation de l'évolution des symptômes sexuels chez les délinquants sexuels atteints de paraphilie (avec ou sans traitements antiandrogènes ou ISRS) »

- ESPARA -

#### RIPH2 - HPS

#### PROTOCOLE DE RECHERCHE

Version n °2.0du 07/02/2025 Réf. promoteur : D24-P008 IDRCB : 2024-A01543-44

Investigateur Coordonnateur

**Professeur Florence THIBAUT** 

Service de Psychiatrie-Addictologie, CHU Cochin

(Groupe Hospitalier APHP.5) Université de Paris Cité

INSERM U1266, Institut de Psychiatrie et

Neurosciences Tél: 01 58 41 16 79

Courriel: florence.thibaut@aphp.fr

Promoteur Groupe Hospitalier Universitaire Paris Psychiatrie &

**Neurosciences (GHU Paris)** 

1, rue Cabanis 75674 Paris Cedex 14

Représenté par Délégation à la Recherche Clinique et à l'Innovation

(DRCI)

1, rue Cabanis 75674 Paris Cedex 14

Structure chargée du suivi de la DRCI

**Recherche** Docteur Khaoussou SYLLA

Coordinateur Médical



# Page de SIGNATURE PROTOCOLE DE RECHERCHE IMPLIQUANT LA PERSONNE HUMAINE

Titre : Etude sur l'observation de l'évolution des symptômes sexuels chez les délinquants sexuels atteints de paraphilie (avec ou sans traitements antiandrogènes ou ISRS).

Version n° 2.0 du : 07/02/2025 IDRCB : 2024-A01543-44

Référence promoteur : D24-P008

La recherche sera conduite conformément au protocole, aux bonnes pratiques en vigueur et aux dispositions législatives et réglementaires en vigueur.

| L'investigateur coordonnateur : Professeur Florence THIBAUT Service de Psychiatrie-Addictologie, CHU Cochin (Groupe Hospitalier APHP.5) Université de Paris Cité INSERM U1266, Institut de Psychiatrie et Neurosciences | Date:///Signature: |
|---|---|
| Le promoteur Son Représentant D.R.C.I. Docteur Khaoussou SYLLA Coordinateur Médical | Date ://// |
| <b>Biostatisticien</b> Madame Rossella Letizia MANCUSI DRCI - GHU Paris | Date ://// |

La recherche a reçu un avis favorable du CPP Est IV en date du 20/mars/2025



# TABLE DES MATIÈRES

| 1 | | RÉSUMÉ SYNOPTIQUE | 5 |
|---|---|---|---|
| 2 | | JUSTIFICATION SCIENTIFIQUE DE LA RECHERCHE | 11 |
| | 2.1<br>2.2<br>2.3<br>2.4<br>2.5 | ETAT ACTUEL DES CONNAISSANCES AU REGARD DE LA RECHERCHE. HYPOTHÈSES DE LA RECHERCHE. DESCRIPTION DE LA POPULATION À ÉTUDIER ET JUSTIFICATION DE SON CHOIX. DESCRIPTION DES ACTES ET DES PROCÉDURES AJOUTÉS PAR LA RECHERCHE. RÉSUMÉ DES BÉNÉFICES ET DES RISQUES PRÉVISIBLES ET CONNUS POUR LES PERSONNES SE PRÊT À LA RECHERCHE. | 12<br>13<br>27 |
| 3 | | OBJECTIFS DE LA RECHERCHE | 29 |
| | 3.1<br>3.2 | OBJECTIF PRINCIPAL DE LA RECHERCHEOBJECTIFS SECONDAIRES DE LA RECHERCHE. | |
| 4 | | CONCEPTION DE LA RECHERCHE | 30 |
| | 4.1<br>4.2<br>4.3 | CRITÈRE D'ÉVALUATION DE LA RECHERCHE | 31 |
| 5 | | DEROULEMENT DE RECHERCHE | 33 |
| | 5.1<br>5.2 | CALENDRIER DE LA RECHERCHE | |
| 6 | | CRITERES D'ELIGIBILITE | 41 |
| | 6.1<br>6.2<br>6.3 | Critères d'inclusion. Critères de non inclusion. Modalités de recrutement. | 41 |
| 7 | | RÈGLES D'ARRÊT | 42 |
| | 7.1<br>7.2<br>7.3 | CRITETRES ET MODALITES D'ARRET PREMATURE DE LA RECHERCHE | 42 |
| 8 | | VIGILANCE | 43 |
| | 8.1<br>8.2 | COMITÉ SPECIQUE DE LA RECHERCHE | |
| 9 | | GESTION DES DONNEES | 43 |
| | 9.1<br>9.2<br>9.3 | MODALITÉS DE RECUEIL DES DONNÉES TRAITEMENT DES DONNÉES ET CONSERVATION DES DOCUMENTS ET DES DONNÉES PROPRIETES DES DONNÉES | 44 |
| 10 | 9.2<br>9.3 | TRAITEMENT DES DONNÉES ET CONSERVATION DES DOCUMENTS ET DES DONNÉES | 44 |
| 10 | 9.2<br>9.3 | TRAITEMENT DES DONNÉES ET CONSERVATION DES DOCUMENTS ET DES DONNÉES | 44<br>45 |



| 11 | CONTRÔLE ET ASSURANCE DE LA QUALITE | 48 |
|---|---|---|
| 11.1 | Organisation générale | |
| 11.2 | STRATEGIE D'OUVERTURE DES CENTRES | 48 |
| 11.3 | CONTRÔLE QUALITE DES DONNEES | |
| 11.4 | CAHIER D'OBSERVATION | |
| 11.5 | GESTION DES NON CONFORMITES | |
| 11.6 | AUDIT | 49 |
| 12 | ASPECTS ETHIQUES ET LEGAUX | 50 |
| 12.1 | MODALITÉS D'INFORMATION ET DE RECUEIL DU CONSENTEMENT DES PERSO | |
| 400 | PRÊTANT A LA RECHERCHE | |
| 12.2 | INTERDICTION POUR LA PERSONNE DE PARTICIPER A UNE RECHERCHE OU I | |
| 10.0 | D'EXCLUSION PRÉVUE A L'ISSUE DE LA RECHERCHE, LE CAS ÉCHÉANT | |
| 12.3 | INDEMNISATION DES SUJETS | |
| 12.4 | OBLIGATIONS LEGALES | 51 |
| 13 | FINANCEMENT ET ASSURANCE | 52 |
| 13.1 | SOURCE DE FINANCEMENT | 52 |
| 13.2 | ASSURANCE | 52 |
| 14 | REGLES RELATIVES A LA PUBLICATION | 52 |
| 14.1 | MENTION DE L4AFFILIATION DU GHU PARIS POUR LES PROJETS PROMUS OU GÉ | ÉRÉS |
| 14.1 | MENTION DE L4AFFILIATION DU GHU PARIS POUR LES PROJETS PROMUS OU GÉ<br>PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & | ÉRÉS |
| 14.1 | · | |
| 14.1<br>14.2 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & | 53 |
| | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES | 53<br>S » DU<br>52 |
| | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES | 53<br>S » DU<br>52 |
| 14.2 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES | 53<br>TS » DU<br>52 |
| 14.2 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES | 53<br>S » DU<br>52<br>S52 |
| 14.2<br>14.3<br><b>15</b> | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES. MENTION DU PROMOTEUR GHU PARIS (DRCI) DANS LES « ACKNOWLEDGMENT MANUSCRIT MENTION DU FINANCEUR DANS LES « ACKNOWLEDGMENTS » DU MANUSCRIT BIBLIOGRAPHIE. | 53 CS » DU52 C5253 CM, |
| 14.2<br>14.3<br><b>15</b> | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES | 53 CS » DU52 C5253 CM, |
| 14.2<br>14.3<br><b>15</b><br>15.1 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES. MENTION DU PROMOTEUR GHU PARIS (DRCI) DANS LES « ACKNOWLEDGMENT MANUSCRIT MENTION DU FINANCEUR DANS LES « ACKNOWLEDGMENTS » DU MANUSCRIT BIBLIOGRAPHIE. ECHELLES D'AGRESSION ET DE VIOL, MOLEST AND RAPE SCALES (Bumby 1996) (Traduction française : T Pham). | 53 CS » DU5253 CM,59 |
| 14.2<br>14.3<br><b>15</b><br>15.1 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES | 53 CS » DU5253 CM,59 |
| 14.2<br>14.3<br>15<br>15.1<br>15.2 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES. MENTION DU PROMOTEUR GHU PARIS (DRCI) DANS LES « ACKNOWLEDGMENT MANUSCRIT MENTION DU FINANCEUR DANS LES « ACKNOWLEDGMENTS » DU MANUSCRIT BIBLIOGRAPHIE ECHELLES D'AGRESSION ET DE VIOL, MOLEST AND RAPE SCALES (Bumby & 1996) (Traduction française : T Pham) L'ECHELLE D'EMPATHIE (BES Basic Empathy Scale) (Joliffe et Farrington., 2006; Traduction française D'Ambrosio et al. 2008) GRILLE D'EVALUATION DU DENI ET DE LA MINIMISATION (McKibben A, Aubut J, Dassylva B (1995). Grille d'évaluation du déni et de la minimisation | 53 CS » DU5253 CM,59 |
| 14.2<br>14.3<br>15<br>15.1<br>15.2 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES. MENTION DU PROMOTEUR GHU PARIS (DRCI) DANS LES « ACKNOWLEDGMENT MANUSCRIT | 53 CS » DU5253 CM,5959 |
| 14.2<br>14.3<br>15<br>15.1<br>15.2<br>15.3<br>15.4 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES. MENTION DU PROMOTEUR GHU PARIS (DRCI) DANS LES « ACKNOWLEDGMENT MANUSCRIT MENTION DU FINANCEUR DANS LES « ACKNOWLEDGMENTS » DU MANUSCRIT BIBLIOGRAPHIE ECHELLES D'AGRESSION ET DE VIOL, MOLEST AND RAPE SCALES (Bumby & 1996) (Traduction française : T Pham) L'ECHELLE D'EMPATHIE (BES Basic Empathy Scale) (Joliffe et Farrington., 2006; Traduction française D'Ambrosio et al. 2008) GRILLE D'EVALUATION DU DENI ET DE LA MINIMISATION (McKibben A, Aubut J, Dassylva B (1995). Grille d'évaluation du déni et de la minimisation QUESTIONNAIRE D'HISTOIRE TRAUMATIQUE, Trauma History Questionnaire (THC (Hooper et al., 2011 traduction française : Jehel et al., 2000) | 53 CS » DU5253 CM,5959 |
| 14.2<br>14.3<br><b>15</b><br>15.1<br>15.2<br>15.3 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES | 53 CS » DU5253 CM,595959 |
| 14.2 14.3 15 15.1 15.2 15.3 15.4 15.5 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES | 53 CS » DU5253 CM,59595959 |
| 14.2<br>14.3<br>15<br>15.1<br>15.2<br>15.3<br>15.4 | PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES | 53 CS » DU5253 CM,5959595959 |



# 1. RÉSUMÉ SYNOPTIQUE

| Titre complet | Etude sur l'observation de l'évolution des symptômes sexuels chez les délinquants sexuels atteints de paraphilie (avec ou sans traitements antiandrogènes ou ISRS) |
|---|---|
| Acronyme/<br>référence | ESPARA / D24-P008 |
| Investigateur<br>coordonnateur | Professeur Florence THIBAUT Service de Psychiatrie-Addictologie, CHU Cochin (Groupe Hospitalier APHP.5) Université de Paris Cité INSERM U1266, Institut de Psychiatrie et Neurosciences Tél: 01 58 41 16 79 Courriel: <a href="mailto:florence.thibaut@aphp.fr">florence.thibaut@aphp.fr</a> |
| Responsable scientifique | Dr Sandrine LAMY |
| Promoteur | Groupe Hospitalier Universitaire - Psychiatrie & Neurosciences (GHU Paris) |
| Justification scientifique | Jusqu'à présent, peu d'études menées sur des petites séries de patients ont été publiées et les connaissances scientifiques sur le traitement des délinquants sexuels paraphiles sont modestes (en particulier concernant l'évaluation des symptômes sexuels chez les patients recevant ou non ces traitements, leurs indications respectives (ISRS et traitements antiandrogènes) et enfin l'observation des effets indésirables). Les recommandations actuelles de prescription des traitements pharmacologiques chez des sujets paraphiles préconisent soit les antidépresseurs sérotoninergiques soit les traitements antiandrogènes en plus du traitement psychologique selon le niveau de gravité du trouble paraphile et le risque de délinquance sexuelle (Recommandations de la Haute Autorité de Santé, 2010 révision 2019; Florence Thibaut, Paul Cosyns, John Paul Fedoroff, Peer Briken, Kris Goethals, John M. W. Bradford & The WFSBP Task Force on Paraphilias (2020) The World Federation of Societies of Biological Psychiatry (WFSBP) 2020 guidelines for the pharmacological treatment of paraphilic disorders, The World Journal of Biological Psychiatry, 21:6, 412-490, DOI: 10.1080/15622975.2020.1744723 En France (ainsi que dans de nombreux pays en Europe), dans un contexte de faibles preuves scientifiques, l'Agence française du médicament a approuvé deux traitements antiandrogènes chez les sujets paraphiles: l'acétate de cyprotérone et la triptoréline. Les ISRS ne sont pas encore approuvés dans le traitement des troubles paraphiles. Néanmoins, les ISRS sont utilisés chez 12% des délinquants sexuels en Allemagne et plus de la moitié des patients aux Etats-Unis sans preuves scientifiques de leur efficacité ou de leur tolérance dans cette indication. Pour des raisons éthiques (risque de victimisation), des études contrôlées randomisées à long terme versus placebo ne sont pas possibles chez des délinquants sexuels ambulatoires. Dans ce contexte, nous souhaitons effectuer une étude naturalistique de suivi prospectif afin d'observer l'évolution des s |
| Objectif | Objectif Principal: |
| principal | Evolution des symptômes sexuels chez les sujets paraphiles inclus dans l'étude (3 groupes de patients : patients sous antiandrogènes, patients sous ISRS et patients sans |



traitements pharmacologiques de type ISRS ou antiandrogène).

# Objectifs Secondaires:

- 1. Estimation du taux de rechute (reprise d'un comportement sexuel déviant) et facteurs associés à la rechute. Les rechutes seront analysées statistiquement si leur nombre est suffisant, mais ne peuvent pas être un objectif prioritaire en raison de leur rareté attendue ;
- 2. Le rôle des troubles psychiatriques concomitants, des troubles de la personnalité et de l'impulsivité dans l'efficacité du traitement, de l'observance (si traitement pharmacologique) et du risque de rechute sera étudié en tenant compte de la gravité et du type de troubles paraphiles ;
- 3. Déterminer les facteurs pouvant être associés à l'évolution des symptômes sexuels, à l'efficacité des traitements et aux effets indésirables potentiels ;
- 4. Analyse des éventuels effets indésirables chez les sujets sous traitements pharmacologiques (ISRS ou antiandrogènes versus sans traitements) ;
- 5. Les modifications des caractéristiques cliniques et cognitives des délinquants sexuels au fil du temps et leurs relations avec l'évolution des symptômes sexuels, l'observance (si traitement pharmacologique) et les risques de rechute seront analysées. En particulier, l'utilisation de pornographie, d'alcool et de drogues illicites, le rôle de l'hypersexualité comorbide et les caractéristiques cognitives telles que : les distorsions cognitives, l'empathie, le déni, seront étudiés dans cette population, en tenant compte de la gravité et du type de troubles paraphiles. La plupart de ces facteurs sont couramment acceptés comme prédicteurs valides de la réponse au traitement, malgré l'absence de recherche systématique pour soutenir ces hypothèses. Le déficit d'évaluation psychométrique pour mesurer ces facteurs contribue aux difficultés de la recherche dans ce domaine. Dans cette étude, nous allons utiliser des échelles d'évaluation spécifiques validées en français pour analyser l'hypersexualité et les caractéristiques cognitives connues pour être associées à la délinquance ;
- 6. Le rôle des trajectoires de vie, avec un focus particulier sur les antécédents de violence physique ou sexuelle et l'exposition à la pornographie durant l'enfance, dans l'efficacité du traitement dans les groupes traités, de l'observance et du risque de rechute sera étudié en tenant compte de la gravité et du type de troubles paraphiles;
- 7. Estimation du nombre de sujets pour qui une modification de la prise en charge est proposée au cours de l'étude et analyse épidémiologique de ce groupe en termes de comorbidité, tolérance aux traitements, évolution des symptômes sexuels.

# Critères d'évaluation

<u>Le critère d'évaluation principal</u> est d'évaluer l'évolution des symptômes sexuels (intensité du désir sexuel et échelle de mesure des symptômes de comportement sexuel déviant (auto-évaluation) mesurés tous les 3 mois.

#### Critères d'évaluation secondaires :

1. Les rechutes éventuelles seront évaluées lors des visites trimestrielles : qu'elles soient déclarées lors des entretiens ou connues par d'autres sources (notification par la famille, les soignants, la justice, etc....). Les rechutes seront enregistrées par l'investigateur et immédiatement signalée au coordinateur. En cas d'incarcération, le patient sortira de l'étude.



- 2. Diagnostic de troubles psychiatriques concomitants : critères DSM-5 ; évaluation des troubles de la personnalité : PDQ-4+ (à l'inclusion) ; Impulsivité : BIS 11 (à l'inclusion).
  - Observance du traitement : pour tous les patients échelle abrégée Brief Adherence Rating Scale (BARS). Pour les patients traités à l'ISRS et aux antiandrogènes : la concentration plasmatique de la testostérone sera mesurée à l'inclusion et en cas de doute sur l'observance.
- 3. Facteurs génétiques (\*) : prélèvement salivaire et prélèvement sanguin (le patient devra donner explicitement son consentement pour l'examen génétique).
- 4. Analyse des éventuels effets secondaires signalés par le médecin en charge du patient ou par le patient lui-même : le type, la fréquence, le moment de survenue d'événements indésirables, ainsi que, le cas échéant, la nécessité d'une consultation médicale, d'une hospitalisation, d'un arrêt de travail, de modifications ou d'une interruption du traitement en raison d'effets indésirables, seront recueillis. Ceci nous permettra de comparer les groupes recevant des ISRS ou des antiandrogènes aux non traités.
- 5. L'examen clinique à l'inclusion et tous les 3 mois :
  - Gynécomastie cliniquement observable (présence ou absence), la mesure de la pression artérielle, du poids.
  - Fonctionnement cognitif : échelle d'agression et de viol (MOLEST et RAPE scales) échelle de déni et d'empathie.
  - Questionnaire AUDIT pour l'alcool (autoquestionnaire d'aide au repérage de la consommation excessive). La consommation d'alcool : (grammes d'alcool pur par jour, nombre maximal de verres par occasion et ancienneté de la consommation) (à l'inclusion et à M36).
  - La Consommation de drogues illicites : type et quantité par jour, ancienneté de la consommation sera évaluée (à l'inclusion et tous les 3 mois).
  - Hypersexualité : PATHOS / PEACCE pour le diagnostic ; Compulsive Sexual Behavior Inventory pour l'évaluation d'une hypersexualité si Pathos positive (≥ 3) (à l'inclusion et à M36). Evaluation du risque de violence sexuelle : STABLE 2007 et Static 99 (à l'inclusion et à M 36).
  - Evaluation cognitive (MoCA) et Stroop (à l'inclusion et à M 36).
- 6. Evaluation des trajectoires de vie traumatiques : THQ Les trajectoires de vie traumatisantes seront évaluées à l'inclusion à l'aide de la version française du Questionnaire d'Histoire des Traumatismes (recherche de toutes sortes de traumatisme) (Trauma History Questionnaire (THQ)) (à l'inclusion).
- 7. Les modifications du plan de traitement seront vérifiées et notifiées lors des visites tous les trois mois
- (\*) A l'inclusion, deux prélèvements pour la réalisation d'une étude génétique seront prélevés. Un échantillon salivaire (1 pot plastique spécifique pour étude de génétique dans lequel le prélèvement salivaire sera réalisé, les échantillons salivaires se conservent



| | à l'état ambiant. Ils seront rapatriés vers le centre INSERM U1266 par un transporteur spécialisé. Seront également prélevés deux tubes EDTA 4ml de sang (par un médecin ou une infirmière), ces tubes seront stockés entre -20°C et -80°C. Si un Centre de Ressources biologiques (CRB) est proche du lieu de prélèvement, les tubes sanguins seront stockés au CRB avant d'être acheminés à la fin de la première année d'inclusion vers le centre INSERM U1266 dans le laboratoire où travaille le Pr Thibaut. S'il n'y a pas de CRB proche du lieu de prélèvement, les tubes seront stockés dans un congélateur dédié à cet effet dans le centre d'inclusion. Un transporteur, à la fin des inclusions, sera chargé de faire parvenir l'ensemble des prélèvements au centre INSERM U1266. Une collection biologique sera réalisée avec ces prélèvements. |
|---|---|
| Schéma<br>expérimental | Suivi observationnel de cohorte. |
| Population concernée | Homme délinquant sexuel atteint de paraphilie. |
| Critères<br>d'éligibilité | <ul> <li>Critères d'inclusion:</li> <li>Hommes souffrant de paraphilies (critères DSM-5),</li> <li>Agés de 18 à 65 ans,</li> <li>Délinquants sexuels (délit ou agression à caractère sexuel incluant exhibitionnisme, viol, attouchement sexuel, inceste, détention de matériel vidéo à caractère pédopornographique) (niveau de gravité 1 à 6 selon les recommandations de la WFSBP),</li> <li>Sujet ayant donné son consentement,</li> <li>Patients pris en charge par la sécurité sociale,</li> <li>Maîtrise satisfaisante du français écrit et parlé.</li> <li>Critères de non inclusion:</li> <li>Sujet en prison (quel qu'en soit le motif),</li> <li>Sujet sous mesure de tutelle (les patients sous curatelle pourront en revanche être inclus),</li> <li>Les sujets ayant commis une infraction sexuelle et qui ne répondent pas aux critères DSM-5 de paraphilie.</li> </ul> |
| Actes ou<br>Produit faisant | Evaluation des symptômes sexuels chez les sujets paraphiles pris en charge avec ou sans traitements pharmacologiques |
| l'objet de la<br>recherche | La prescription est indépendante de la recherche, les produits sont utilisés conformément à leur AMM ou aux recommandations professionnelles incluant les recommandations de l'ANSM de juin 2019 concernant l'acétate de cyprotérone. Il n'y aura aucun impact du protocole sur les posologies ou modalités d'administration (la prescription est antérieure à la proposition d'inclure le patient dans la recherche et indépendante de celle-ci. De même, l'évolution de la prescription pendant la période de participation indépendante du protocole relève exclusivement de la décision du praticien suivant chaque patient). |
| Autres actes<br>ou procédures<br>ajoutés par la<br>recherche | La recherche se propose de systématiser la surveillance clinique et biologique conforme aux bonnes pratiques lors de la prise en charge pharmacologique et psychologique des sujets paraphiles. Des évaluations psychologiques et psychiatriques complémentaires sont prévues sous forme d'échelles et de questionnaires autorapportés. Une recherche génétique est également prévue (le patient devra donner explicitement son consentement pour l'examen génétique). |



| Bénéfices<br>attendus pour | À notre connaissance, cette cohorte sera la plus grande population de délinquants sexuels |
|---|---|
| | paraphiles étudiés pendant la durée la plus longue à ce jour dans un champ où la |
| les | recherche est insuffisante. |
| participants et | Ce vaste échantillon bénéficiant de soins de routine et suivis pendant 3 ans va nous |
| pour la société | permettre d'analyser l'évolution des patients selon la prise en charge reçue par leur |
| pour lu societe | psychiatre traitant. |
| Risques et | La systématisation du recueil d'événements et de la surveillance des effets des |
| contraintes | traitements ne constitue pas un risque supplémentaire par rapport à un suivi habituel. |
| minimes | L'ostéodensitométrie fait partie des examens complémentaires envisagés lors d'un suivi |
| ajoutés par la | classique, l'irradiation est très faible, moindre que pour une radiologie classique. |
| recherche | Il n'y a pas de risque attendu avec les prélèvements. Les outils d'évaluation |
| | psychologique utilisés sont des outils cliniques classiques. Leur passation sera réalisée |
| | dans un contexte d'examen médical et paramédical, ce qui permettra la reprise |
| | d'éléments émergents éventuels avec le praticien. |
| | Au total, le risque peut être considéré comme minime. |
| Déroulement | Après information et recueil du consentement, les patients traités par antiandrogènes ou |
| pratique | ISRS ou aucun des deux seront inclus de manière naturalistique, sans que l'inclusion |
| pranque | n'influence la prise en charge thérapeutique. Les sujets seront inclus sur leur lieu de soin |
| | habituel. Ils bénéficieront d'une évaluation complète médicale et paramédicale, |
| | psychiatrique et psychologique à l'inclusion. Des autoquestionnaires permettant de |
| | mieux appréhender leur fonctionnement ainsi que des outils d'évaluation des |
| | symptômes sexuels et du risque de récidive seront évalués sur dossier. |
| | Durant une période de 3 ans, ils seront suivis tous les 3 mois, avec évaluation du suivi, de |
| | l'observance, recueil des événements indésirables et de paramètres cliniques évaluant les |
| | symptômes sexuels et la tolérance des traitements dans les groupes où ils sont présents. |
| | Lors de la visite finale, l'évaluation comprendra outre les paramètres recueillis lors du |
| | suivi une évaluation biologique identique à l'évaluation initiale. Les prélèvements |
| | destinés à l'étude génétique seront réalisés à l'inclusion. |
| | Une collection biologique sera réalisée à partir de ces prélèvements. |
| Nombre de | |
| | Il est prévu d'inclure 200 hommes délinquants sexuels paraphiles. On en attend environ |
| sujets | 100 recevant des traitements pharmacologiques (ISRS ou anti-androgènes): 75 dans le groupe ISRS, et 25 (correspondant à 100 personnes-années) dans le groupe traité par |
| | antiandrogènes, et environ 100 dans le groupe sans ISRS et sans antiandrogènes. |
| Centres | <u> </u> |
| Investigateurs | Recherche multicentrique nationale |
| Calendrier de | Durée d'inclusion : 24 mois |
| la recherche | Durée de participation des patients (traitement + suivi) : 3 ans |
| | > Durée totale : 5 ans |
| Analyse | Des analyses distinctes seront conduites dans chacun des trois groupes (patients |
| statistique | recevant des ISRS, patients recevant des anti-androgènes et patients ne recevant aucun de |
| | ces traitements). Si les caractéristiques des différents groupes le permettent, des |
| | comparaisons entre ces groupes seront réalisées après ajustement sur les caractéristiques |
| | des sujets. |
| | Les principaux critères d'évaluation seront les scores de l'intensité du désir sexuel (libido |
| | et désir, des pensées sexuelles ou fantasmes, l'activité sexuelle). De plus, les scores seront |
| | dichotomisés, séparant les sujets sans intérêt sexuel paraphile, pas de pensées ou pas |
| | arctiotoffices, separati les sujets suits interet sexuer paraprine, pas de perisces ou pas |
| | d'activité (score étant égal à 0), résultat qui peut être considéré comme définissant un |
| Calendrier de<br>la recherche<br>Analyse | <ul> <li>Durée d'inclusion : 24 mois</li> <li>Durée de participation des patients (traitement + suivi) : 3 ans</li> <li>Durée totale : 5 ans</li> <li>Des analyses distinctes seront conduites dans chacun des trois groupes (patients recevant des ISRS, patients recevant des anti-androgènes et patients ne recevant aucun de ces traitements). Si les caractéristiques des différents groupes le permettent, des comparaisons entre ces groupes seront réalisées après ajustement sur les caractéristiques</li> </ul> |



| | courante permettront d'évaluer les évènements indésirables s'ils sont observés. D'autres analyses examineront les scores de l'intensité du désir sexuel et de rechute des infractions sexuelles. |
|---|---|
| | Des modèles multivariés seront construits afin de déterminer les caractéristiques associées de façon indépendante avec les résultats, avec la possibilité d'inclure des caractéristiques variables dans le temps, permettant des observations répétées au cours du suivi. Tous les tests seront bilatéraux et 5% sera choisi comme niveau de significativité. Comité de surveillance : aucun (étude d'observation de prescriptions habituelles, pas de risque supplémentaire lié à l'étude attendu). |
| Source de financement | PHRC National 2015 |



# 2. <u>JUSTIFICATION SCIENTIFIQUE DE LA RECHERCHE</u>

#### 2.1 ETAT ACTUEL DES CONNAISSANCES AU REGARD DE LA RECHERCHE

# 2.1.1 Sur la pathologie

En France, le nombre d'agressions sexuelles continue d'augmenter + 20% au cours des 5 dernières années ; environ 33 plaintes pour viols sont enregistrées par jour selon l'Observatoire National de la Délinquance (données communiquées par la gendarmerie Nationale, www.inhesj.fr). Dans l'enquête CIASE 2020, 19.2% des femmes et 7.9% des hommes de 18 à 69 ans rapportent avoir subi des violences sexuelles au cours de leur vie (dont 40% de viols) (28,010 personnes interrogées à distance anonymement par IPSOS) ; 95% des agresseurs sont des hommes (un inconnu dans la rue dans seulement 15% des cas ; dans les autres cas l'agresseur était connu de la victime ou de la famille au préalable) et plus de 70% des victimes l'ont été avant l'âge de 18 ans. Or, seulement 13% des victimes portent plainte et au final seulement 35% des agresseurs ayant fait l'objet d'une plainte sont condamnés.

Les conséquences personnelles et sociales des viols et violences sexuelles sont pourtant un problème majeur de santé publique (Felitti, 1991; Thibaut 2015); 90-95% des victimes ont des conséquences psychologiques et/ou physiques selon un rapport européen (<a href="https://www.europeanceo.com/business-and-management/the-cost-of-sexual-assault/">https://www.europeanceo.com/business-and-management/the-cost-of-sexual-assault/</a>). Le coût annuel des violences sexuelles est estimé à 1.5 à 2% du produit intérieur brut soit environ 35 euros par habitant par an (<a href="https://www.europeanceo.com/business-and-management/the-cost-of-sexual-assault/">https://www.europeanceo.com/business-and-management/the-cost-of-sexual-assault/</a>).

Tous les auteurs sont d'accord pour dire que l'incarcération seule ne résout pas le problème de la violence sexuelle et que le traitement médical des délinquants sexuels est une étape critique dans la prévention de la récidive, en particulier chez les personnes à risque élevé de violence comme les pédophiles et les violeurs récidivistes (Garcia et Thibaut, 2011; Thibaut, 2013).

# 2.1.2 Sur les stratégies/procédures de référence

Malheureusement, en dépit de l'utilisation croissante des traitements pharmacologiques dans ces indications, nous disposons de peu de données pour indiquer quelles populations de délinquants sexuels pourront bénéficier de quels traitements pharmacologiques et avec quelle efficacité, quels événements indésirables sont observés, en particulier avec les anti-androgènes ou les traitements antidépresseurs qui sont largement utilisés chez ces sujets. Une étude Cochrane a montré que le traitement psychodynamique est moins efficace en termes de délinquance sexuelle par rapport à la probation seule et n'a pas montré d'efficacité significative de la thérapie cognitivocomportementale (TCC) par rapport à l'absence de traitement, sauf pour une étude dans laquelle le traitement anti-androgène a été associé à la TCC (Dennis et al., revue Cochrane 2012). Une autre analyse Cochrane (Khan et al. 2015) a conclu que la tolérance, même des médicaments antiandrogènes, était incertaine étant donné que toutes les études étaient de petite taille et de durée limitée et que de nouvelles recherches étaient nécessaires en utilisant des échantillons plus importants, une durée plus longue du traitement et l'évaluation des médicaments les plus souvent utilisés (en particulier les ISRS ou les analogues de la GnRH). Néanmoins, dans ce contexte de faibles preuves scientifiques, les ISRS ont été utilisés dans la moitié des programmes communautaires en Allemagne et en Amérique du Nord sans preuves scientifiques d'efficacité dans cette indication (Mc Grath et al., 2010). L'acétate de cyprotérone a été approuvé pour la



« modération de désir sexuel chez les hommes adultes atteints de déviance sexuelle » (Androcur® 100mg) (07/2005) et la triptoréline (Salvacyl®, 11,25 mg action prolongée formulation im) pour "diminution réversible des taux de testostérone jusqu'à des niveaux de castration afin de diminuer le désir sexuel chez les hommes adultes atteints de déviance sexuelle "(08/2007). La "Haute Autorité de Santé" et la Fédération mondiale des sociétés de psychiatrie biologique (WFSBP) ont publié des recommandations concernant le traitement pharmacologique des paraphilies (HAS 2010 ; Thibaut et al., 2020).

Par conséquent, il est essentiel de procéder à une vaste étude prospective et de suivi longitudinal dans des conditions naturalistiques dans cette population de délinquants sexuels paraphiles afin d'évaluer l'évolution des symptômes sexuels chez les sujets en fonction de la prise en charge (avec ou sans traitement pharmacologique). Cette étude sera cruciale afin d'améliorer nos connaissances dans le domaine du suivi des délinquants sexuels.

#### 2.2 HYPOTHESES DE LA RECHERHCE

À notre connaissance, cette cohorte sera la plus grande population de délinquants sexuels paraphiles étudiés pendant la durée la plus longue à ce jour dans un champ où la recherche est insuffisante.

Ce vaste échantillon bénéficiant de soins de routine et suivis pendant 3 ans va nous permettre d'analyser l'évolution des patients selon la prise en charge reçue par leur psychiatre traitant.

En outre, cette analyse des pratiques cliniques sera cruciale pour améliorer nos connaissances sur les indications de ces traitements, qui pourraient éventuellement être revues en ce qui concerne leur efficacité et la tolérance, en particulier dans les cas les plus graves de délinquants sexuels avec paraphilie.

Une analyse Cochrane (Khan et al. 2015) a conclu (1) que la tolérance des traitements était incertaine étant donné que toutes les études étaient de petite taille (et donc de faible puissance pour évaluer les effets défavorables) et d'une durée limitée, qui ne correspond pas à la pratique actuelle de routine clinique (surtout chez les jeunes sujets suivis pendant plusieurs années) et (2) que des recherches supplémentaires sont nécessaires devant inclure des tailles d'échantillons plus grands sur de plus longues durées de suivi.

Parallèlement à l'éducation des enfants et au diagnostic, et à la prise en charge précoce des victimes de violence sexuelle, le traitement des délinquants sexuels est un élément clé dans la réduction de la violence sexuelle et de ses conséquences graves sur les victimes en particulier pour les délinquants sexuels les plus graves (sujets pédophiles et violeurs en série) (Gene et al, 2001; Thibaut F. Approche psychiatrique des Déviances Sexuelles Ed Springer Verlag, 2013; Hanson et al, 2014; Thibaut F. Abus Ed O Jacob 2015). Un rapport estime que l'abus sexuel des enfants a coûté 6.7 milliards d'euros en 2018-2019 au Royaume-Uni (seulement pour la prise en charge des victimes) (<a href="https://www.gov.uk/government/publications/the-economic-and-social-cost-of-contact-child-sexual-abuse/the-economic-and-social-cost-of-contact-child-sexual-abuse/the-economic-and-social-cost-of-contact-child-sexual-abuse).

La systématisation du recueil d'événements et de la surveillance des effets des traitements ne constitue pas un risque supplémentaire par rapport à un suivi habituel. L'ostéodensitométrie fait partie des examens complémentaires envisagés lors d'un suivi classique, l'irradiation est très faible, moindre que pour une radiologie classique. Il n'y a pas de risque attendu avec les prélèvements. Les outils d'évaluation psychologique utilisés sont des outils cliniques classiques. Leur passation sera réalisée dans un contexte d'examen médical, ce qui permettra la reprise d'éléments émergents éventuels avec le praticien.

Au total, le risque peut être considéré comme minime.



# 2.3 DESCRIPTION DE LA POPULATION A ETUDIER ET JUSTIFICATION DE SON CHOIX

Dans toutes les formes d'agression sexuelle, une condition nécessaire est que la victime n'ait pas consenti aux gestes sexuels commis, qu'elle était incapable d'y consentir ou de les refuser, ou encore qu'elle n'avait pas l'âge de consentir (par exemple le viol ou l'agression sexuelle, une relation sexuelle incestueuse, une exposition indécente ou exhibition sur des mineurs...). Tous les délinquants sexuels n'ont pas un diagnostic de trouble paraphilique. En fait, il est difficile d'estimer la véritable prévalence des troubles paraphiles dans la population générale car tous les sujets paraphiles ne deviennent pas délinquants sexuels. Étant donné que seuls quelques personnes souffrant de troubles paraphiles, à risque de délinquance sexuelle, demandent volontairement un traitement, la plupart des données disponibles sont basées sur des patients paraphiles ayant été condamnés (Abel et Osborn, 1992; Fagan et al 2002; Hall et Hall, 2007).

# 2.3.1 Epidémiologie:

En France en 2010 (Observatoire International des Prisons, 2010), 14% des 61 000 prisonniers étaient des délinquants sexuels (environ 2% étaient des femmes). Viol et agression sexuelle de femmes constituaient de loin la majorité des infractions sexuelles (dans 72% des cas, la victime avait moins de 18 ans) et la prévalence des agressions sexuelles contre les enfants est en augmentation. On estime qu'à ce jour en France environ 1000 délinquants sexuels sont concernés par une mesure de soins pénalement ordonnés suivant leur incarcération, dont la durée peut varier. Toutefois, aucune donnée nationale n'est disponible dans ce domaine.

Dans notre échantillon régional de 100 délinquants sexuels soumis à des soins pénalement obligés (tout type de traitement) (Haute-Normandie) (99% des hommes, 60% d'agressions sexuelles sur mineurs, 14% d'outrage à la pudeur), un diagnostic de trouble paraphile était posé dans 19% des cas (pédophilie dans 10 cas et exhibitionnisme dans 9 cas respectivement) (Tesson et al. 2012). Dans cette dernière population, le risque de récidive est élevé.

En France, nous avions déjà identifié 345 délinquants sexuels avec des troubles paraphiles entre 2010 et 2014.

# Définition de la paraphilie, comorbidités :

Les paraphilies (à partir de « para » du grec signifiant autour ou à côté et "philos" qui signifie amour) sont des comportements sexuels, des fantasmes ou des actes qui sont déviants par rapport aux comportements sexuels socialement acceptés, mais qui sont nécessaires, et dans certains cas suffisants, pour certaines personnes, à l'obtention d'une excitation sexuelle ou d'un orgasme (Garcia et Thibaut, 2010 ; Thibaut et al, 2013 et 2020).

Le DSM-5 a classé ces troubles de la préférence sexuelle dans le chapitre "Paraphilies" (https://www.psychiatry.org/File%20Library/Psychiatrists/Practice/DSM/APA\_DSM-5-Paraphilic-Disorders.pdf). Le DSM-5, comparativement aux versions antérieures du DSM, a introduit une distinction entre les paraphilies et les troubles paraphiliques "une paraphilie en tant que telle ne justifiant pas systématiquement une intervention psychiatrique et n'étant pas obligatoirement synonyme de trouble paraphilique". Le DSM-5 donne une définition générale des troubles paraphiliques : "Les caractéristiques essentielles d'une paraphilie sont des fantaisies imaginatives sexuellement excitantes, des impulsions sexuelles ou des comportements survenant de façon répétée et intense, et impliquant (i) des objets inanimés, (ii) la souffrance ou l'humiliation de soimême ou du partenaire, (iii) des enfants ou d'autres personnes non consentantes, et qui s'étendent sur une période d'au moins six mois (critère A). Chez certaines personnes, des fantaisies imaginatives (fantasmes) ou des stimuli paraphiliques sont obligatoires pour déclencher une excitation sexuelle et font toujours partie de l'acte sexuel. Chez d'autres, les préférences



paraphiliques n'apparaissent qu'épisodiquement (par exemple au cours de périodes de stress) alors qu'à d'autres moments, la personne est capable d'avoir un fonctionnement sexuel sans faire appel à des fantaisies imaginatives ou à des stimuli paraphiliques. Les comportements, impulsions sexuelles, ou fantaisies imaginatives sont à l'origine d'un désarroi cliniquement significatif ou d'une altération du fonctionnement social, professionnel ou dans d'autres domaines importants (critère B)". Dans le trouble paraphilique, la personne a mis en acte ses besoins sexuels atypiques ou encore ses besoins et fantasmes lui causent une souffrance ou des difficultés interpersonnelles (Thibaut, EMC 2020: Thibaut F. Troubles des conduites sexuelles (troubles paraphiliques) : diagnostic et traitement. EMC - Psychiatrie 2020;36(3):1-15 [Article 37-510-A-50].).

Dans cette conception, avoir une paraphilie serait une condition nécessaire mais pas une condition suffisante pour déterminer l'existence d'un trouble paraphilique. Les troubles paraphiles se sont pas illégaux en eux-mêmes, mais le fait d'agir en réponse à des pulsions paraphiles peut être illégal (infraction sexuelle) et, dans certains cas, pourrait entraîner des sanctions juridiques graves comme fréquemment observé dans le cas de la pédophilie. Les patients souffrant de troubles paraphiles graves viennent généralement consulter après avoir commis un acte sexuel sur un enfant ou un adulte non-consentant. En fait, la plupart d'entre eux ne trouvent pas leurs fantasmes suffisamment stressants ou ego-dystoniques pour demander une prise en charge ou ils peuvent se sentir honteux et ne pas oser demander un avis médical.

Pour certaines personnes (troubles paraphiles exclusifs), les fantasmes ou les stimuli paraphiles sont obligatoires pour obtenir une excitation sexuelle et sont toujours inclus dans leur activité sexuelle. Dans d'autres cas, les préférences paraphiles ne se produisent qu'épisodiquement alors que, à d'autres moments, la personne est capable de fonctionner sexuellement sans la présence de stimuli ou fantasmes déviants.

Le trouble paraphilique est principalement observé chez les hommes (90-99% des cas, sauf pour le masochisme), même si des cas ont été rapportés chez des femmes (moins de 1% des cas) (Maletzki, 1994). Les troubles de l'humeur, les consommations d'alcool ou de toxiques et les troubles anxieux sont les comorbidités les plus fréquemment associées à des troubles paraphiles, avec une prévalence estimée à 61-81%, 50-83% et 31-64% respectivement (Raymond et al 1999;. Galli et al, 1999; McElroy et al, 1999). Le trouble du contrôle des impulsions et le syndrome de stress posttraumatique sont également décrits en association avec des troubles paraphiles (Raymond et al, 2003). Des troubles de la personnalité sont aussi fréquemment observés chez les sujets paraphiles (33-52%) (troubles de la personnalité de type états limites ou antisociaux dans la plupart des cas). Environ 30 à 40% d'entre eux ont été victimes d'abus sexuels et/ou physiques dans l'enfance, en particulier pour les pédophiles (Thibaut, 2013 et 2024 (article soumis)). Une étude récente finlandaise (Alanko et al., 2010) rapporte la contribution de facteurs génétiques dans la pédophilie pouvant expliquer 15% de la variance dans une population de 3,968 jumeaux de sexe masculin. Dans notre population, les rôles respectifs des facteurs environnementaux et génétiques dans les comportements paraphiles pourront ainsi être étudiés puisque nous aurons des informations sur les violences subies dans l'enfance et sur les antécédents personnels et familiaux des patients inclus. Aucune étude épigénétique (études des modifications dynamiques de la régulation des gènes) n'a été menée à ce jour dans ces populations. Or, l'épigénétique joue un rôle important dans l'apparition de troubles psychiatriques et dans le développement sexuel normal et constitue une voie de recherche très prometteuse dans la compréhension des troubles paraphiles (Nugent et al., 2011; Schroeder et al., 2012; Thibaut et al. 2020).



# Évolution et facteurs pronostiques :

Les informations disponibles, concernant l'évolution clinique et les facteurs pronostiques des troubles paraphiles, sont limitées. Une étude réalisée dans une large population de sujets paraphiles ayant agressé sexuellement des enfants a montré que la pédophilie commence tôt : près de 20% des patients atteints de pédophilie ont fait une première victime avant l'âge de 10 ans, 43% a commencé à agresser entre les âges de 10 à 15 et environ 80% d'entre eux déclarent qu'ils ont eu leur premier enfant victime avant l'âge de 20 ans (Abel et Harlow, 2001). La pédophilie est considérée comme un trouble chronique (Murray, 2000; Dickey et al, 2002). Les pédophiles peuvent récidiver à un âge plus élevé comparativement aux autres délinquants sexuels dans une population de 44% de pédophiles parmi les 168 délinquants sexuels âgés de 40 à 70 ans (Dickey et al, 2002). En outre, de 30 à 70% des pédophiles présentent un autre trouble paraphilique (par exemple, un tiers des pédophiles sont également exhibitionnistes) (Abel et al 1988; Raymond et al 1999; Bradford et al, 1992; Galli et al, 1999).

La récidive est un problème majeur durant le traitement de sujets paraphiles. Trois méta-analyses ont décrit les taux de récidive et les facteurs de risque (Craig et al 2008; Hanson et al, 2003; Hanson et Morton-Bourgon, 2005). Le taux de récidive est passé de 15% à 5 ans de 27% à 20 ans de suivi. Les pédophiles attirés par les garçons sont plus susceptibles de récidiver par rapport à ceux attirés par les filles et à ceux qui ont agressé au sein de leur famille (Harris et Hanson, 2004). Chez les adultes (61 études de suivi), Hanson et Bussière (1998) ont rapporté un taux de récidive sexuelle de 13,4% (23 393 cas). Chez les adultes, la récidive sexuelle est surtout prédite par le type de déviance sexuelle et, dans une moindre mesure, par des facteurs généraux criminologiques (âge, nombre d'infractions antérieures, comorbidité psychiatrique, troubles de la personnalité, consommation d'alcool ou toxicomanie) (pour revue voir HAS 2010 et les 2 tableaux ci-dessous) et, surtout une mauvaise observance du traitement. Alexander (1999) a analysé à partir de 79 études publiées entre 1943 et 1996, les résultats des traitements chez 10 988 délinquants sexuels; les analyses basées sur le lieu dans lequel a été conduit le traitement montrent des taux de récidive proches (taux basé sur le nombre de nouvelles arrestations) quelle que soit la localisation (6,3 à 8,5%) (ambulatoire, prison, hôpital ou indéterminée). Les taux de récidive étaient respectivement de 5,8% pour les violeurs et 2,1% pour les agresseurs sexuels d'enfants. Il apparaît ainsi que le traitement des délinquants est essentiel pour prévenir la violence sexuelle et réduire la victimisation.

La relation entre l'hypersexualité, qui est fréquemment associée à des troubles paraphiles, et la délinquance sexuelle doit être étudiée avec soin. L'hypersexualité appelée également comportement sexuel compulsif est définie comme un syndrome clinique caractérisé par des pulsions et comportements sexuels intenses, pénibles et récurrents qui interfèrent avec le fonctionnement quotidien d'une personne. En dépit du désir de se libérer de leurs symptômes, les personnes ayant un comportement sexuel compulsif sont incapables de contrôler leurs comportements et pensées sexuelles pénibles (pour revue Chagraoui et Thibaut, 2016).



| | Facteurs de risque statiques de récidive d'agression sexuelle | | | | |
|---|---|---|---|---|---|
| | Opérationnalisation de la récidive | | | | |
| Types de<br>facteur de<br>risque | Récidive sexue | lle | Récidive non<br>sexuelle | Récidive en généra | |
| Facteurs de Psychopathie risque | | | Psychopathie | Psychopathie | Psychopathie |
| statiques | Agressions sexuelles antérieures | | Agressions sexuelles antérieures | Agressions sexuelles antérieures | Agressions sexuelles antérieures |
| | Déviance sexuelle | | Déviance sexuelle | Déviance sexuelle | |
| | Statut marital (vivre seul) | € | | | Statut marital (vivre seul) |
| | Victime d'abus dan<br>l'enfance | ıs | Antécédents Antécédents familiaux Age jeune familiaux de violence de violence et d'abus physiques | | |
| | Victimes<br>extrafamiliales (noi<br>connues, connues | | | | |
| | | s de | risque dynam | iques de récidi | ve de l'agression |
| sexuell | е | | | | |
| Types de<br>risque | facteur de | Op | pérationnalisatio | on de la récidive : | Récidive sexuelle |
| Facteurs dynamiqu | • | Incapacité à se contrôler | | | |
| | | Со | ngruence émotionr | nelle avec les enfants | 5 |
| | | Colère, Hostilité | | | |
| | | Tendance à se rappeler les émotions négatives | | | |
| | | Faible estime de soi | | | |
| | | Intérêt sexuel inapproprié | | | |
| | | Pré | eoccupations sexue | elles | |
| | | Pe | rsonnalité antisocia | ile | |
| | | Ins | tabilité au travail | | |
| | | Abus et dépendance de substances psycho-actives | | | |
| | | Comorbidités psychiatriques (troubles de la personnalité, psychose) | | | |
| | | Justification des relations sexuelle avec les enfants | | | |
| | | Inc | Incapacité à planifier ses activités personnelles | | |
| | | Ma | Manque de motivation au changement | | |
| | | Adhésion au traitement | | | |



#### 2.3.2 Traitements

La psychothérapie est utilisée chez tous les délinquants sexuels (dans la plupart des cas, la thérapie comportementale est préférée) (Hall et Hall, 2007). Chez les sujets paraphiles à risque élevé de récidive, le traitement pharmacologique devrait être utilisé comme traitement de première intention. Selon les recommandations actuelles, les traitements pharmacologiques comprennent les Inhibiteurs Spécifiques de Recapture de la Sérotonine (ISRS) et les traitements antiandrogènes.

# • ISRS

#### **Efficacité**

La justification de l'utilisation des antidépresseurs sérotoninergiques chez les délinquants sexuels est basée sur plusieurs sources de données (pour revue Thibaut et al, 2010; Assumpçao et al, 2014): (1) dans des modèles animaux, l'augmentation des niveaux de sérotonine dans l'hypothalamus inhibe la motivation sexuelle et la testostérone tandis que l'augmentation des niveaux de sérotonine dans le cortex préfrontal améliore la résilience émotionnelle et le contrôle des impulsions; (2) l'observation clinique des similitudes entre les fantasmes et comportements paraphiles et certains types de symptômes obsessionnels compulsifs; (3) les relations observées entre la dérégulation sérotoninergique et des dimensions spécifiques de la psychopathologie observée dans les troubles paraphiles: impulsivité, comportement antisocial, anxiété, dépression et hypersexualité; et (4) enfin, une meilleure connaissance des effets indésirables des ISRS sur le comportement sexuel, ont suggéré l'utilisation de ces effets indésirables pour le traitement de la déviance sexuelle. En effet, un médicament qui augmente la transmission sérotoninergique centrale a été à l'origine d'une réduction des fantasmes et comportements paraphilies (Jacobsen, 1992).

L'efficacité des ISRS et les effets indésirables observés avec la clomipramine ont limité son utilisation dans le traitement des troubles paraphiles. Dans une revue systématique des données disponibles sur l'efficacité des ISRS dans le traitement des délinquants sexuels, les ISRS ont montré une bonne efficacité clinique pour le traitement des agresseurs sexuels bien que la qualité des études disponibles soit limitée par des biais méthodologiques (par exemple durée de suivi insuffisante, échantillons hétérogènes). Les patients présentant un exhibitionnisme, une masturbation compulsive ou une pédophilie sans passage à l'acte sont des indications d'un traitement par ISRS (Adi, méta-analyse, 2002). L'observance et l'acceptation des ISRS semblent être plus élevées comparativement aux traitements hormonaux chez les délinquants sexuels (Fedoroff, 1995). Plusieurs études ouvertes réalisées avec des ISRS ont montré une diminution des comportements de délinquance sexuelle à court terme. Cependant aucune étude à long terme contrôlée randomisée concernant l'efficacité des ISRS dans le traitement des troubles paraphiles n'a été publiée à ce jour. La fluoxétine et la sertraline ont été les ISRS les plus étudiés dans le traitement des troubles paraphiles. La plupart des données disponibles sont des études de cas et une revue systématique concernant l'utilisation des ISRS chez les délinquants sexuels a retenu seulement neuf séries de cas pour l'analyse (Adi et al., 2002). L'efficacité de la fluoxétine dans la réduction des fantasmes et des comportements paraphiles a été décrite pour le traitement de la pédophilie (Aguierre, 1999; Greenberg et al 1996;. Bourgeois et Klein, 1996; Coleman et al 1992;. Perilstein, 1991), de l'exhibitionnisme (Coleman et al 1992;. Perilstein, 1991; Bianchi, 1990; Yang et Liang, 2010), et des troubles paraphiles en général (Fedoroff, 1995; Greenberg et al 1996; Kafka, 1991,1994; Kafka et Prentky, 1992; Kafka et Hennen, 2000; Galli et al, 1998). Une réponse thérapeutique insuffisante ou nulle avec la fluoxétine a été décrite dans une étude rétrospective portant sur des patients atteints de troubles paraphiles (Bradford et al, 1996) et une étude de cas



concernant un exhibitionniste et un autre avec sadisme sexuel (Wawrose et Sisto, 1992). Quatre essais en ouvert concernant l'utilisation de la fluoxétine chez les patients souffrant de troubles paraphiles ont été publiés. Kafka et Prentky (1992) a traité 10 patients atteints de troubles paraphiles et 10 patients atteints d'hypersexualité et obtenu une réduction significative du comportement sexuel non conventionnel. Un deuxième essai a obtenu 70% de rémission des troubles paraphiles (n = 13) et des troubles liés à la paraphilie (n = 11) après un programme de traitement en deux étapes avec la sertraline suivie par la fluoxétine (Kafka, 1994). Fedoroff et al. (1995) ont obtenu près de 95% de rémission des symptômes avec la fluoxétine en association avec une psychothérapie comparativement à la psychothérapie seule (n = 51). Un dernier essai a obtenu une réduction du nombre total d'actes sexuels et du temps passé dans les comportements paraphiles avec une association de fluoxétine et de méthylphénidate (n = 26) (Kafka, 1994). La stratégie la plus fréquemment utilisée est la titration de la dose jusqu'à l'obtention d'une réduction importante ou la disparition compète des symptômes. La dose moyenne utilisée dans ces études était de 40 mg (20-80) et la durée maximale de traitement était de 4 à 6 semaines. Des études portant sur l'efficacité de la sertraline dans le traitement de la pédophilie (Bradford et al 2000;. Chow et Choy, 2002), des troubles paraphiles (Kafka, 1994; Kafka et Hennen, 2000) et des troubles en lien avec les paraphilies (Kafka, 1994) ont été publiées. Une étude en ouvert de 12 semaines avec titration des doses de sertraline dans le traitement de la pédophilie (n = 20) a montré des réductions des pulsions sexuelles, des fantasmes sexuels, et des comportements sexuels. Ces auteurs ont rapporté une réduction de l'excitation sexuelle avec la suppression de l'excitation déviante, mais un maintien ou une augmentation relative de l'excitation non-pédophile et des relations sexuelles avec des adultes consentants (Bradford, 2000). Une étude rétrospective portant sur 25 patients traités par la sertraline pour pédophilie ou des troubles paraphiles a montré une diminution significative des fantasmes paraphiles (Greenberg et al., 1996). Une autre étude en ouvert a décrit 50% de rémission des symptômes paraphiles en utilisant 100 mg de sertraline pendant une durée moyenne de suivi de 17 semaines (Kafka, 1994). L'efficacité de la fluvoxamine a été décrite chez 16 patients pédophiles (Greenberg et al., 1996) et un patient exhibitionniste avec masturbation compulsive (Zohar et al., 1994). La fluvoxamine a également été associée avec le méthylphénidate et a montré une efficacité dans le traitement de troubles paraphiliques (Kafka et Hennen, 2000).

# Effets indésirables des ISRS:

La majorité des gens n'éprouvent que quelques effets indésirables légers avec les ISRS. Quelquesuns des principaux effets indésirables des ISRS sont décrits ci-dessous, mais cela ne constitue pas une liste exhaustive (National Health Service, Royaume-Uni, www.nhs.uk). Les effets indésirables courants des ISRS peuvent inclure: sensation d'agitation, tremblements ou anxiété, nausées ou vomissements, indigestion, diarrhée ou constipation, perte d'appétit et perte de poids, vertiges, vision floue, bouche sèche, transpiration excessive, insomnie ou somnolence, maux de tête, baisse de la libido, difficulté à atteindre l'orgasme pendant les rapports sexuels ou la masturbation, et chez les hommes difficulté à obtenir ou à maintenir une érection (dysfonction érectile). Des effets indésirables moins communs des ISRS peuvent inclure : des ecchymoses ou des saignements, y compris des vomissements de sang ou la présence de sang dans les selles, une confusion, une rigidité ou des tremblements, des hallucinations visuelles ou auditives, des difficultés à uriner. Le syndrome sérotoninergique est un syndrome rare mais potentiellement grave pouvant survenir avec les ISRS. Il est généralement déclenché quand un ISRS est utilisé en association avec d'autres médicaments (ou substances) qui augmentent également les niveaux de sérotonine, comme un autre antidépresseur, du lithium ou du millepertuis. Les symptômes du syndrome sérotoninergique peuvent inclure : une confusion, une agitation, des spasmes musculaires, des



sueurs, des frissons, de la diarrhée. Les symptômes du syndrome sérotoninergique dans sa forme grave comprennent : une température élevée (fièvre), des convulsions, une arythmie, une perte de conscience. Les personnes âgées qui prennent des ISRS peuvent présenter une hyponatrémie. Une hyponatrémie légère peut provoquer des symptômes similaires à la dépression ou aux effets indésirables des ISRS, tels que : nausées, maux de tête, douleurs musculaires, diminution de l'appétit, confusion. Une hyponatrémie plus sévère peut provoquer les symptômes suivants : sensation apathique et fatigue, une désorientation, une agitation, des symptômes psychotiques, des convulsions, une perte de conscience.

Les jeunes de moins de 25 semblent plus à risque de survenue d'idées ou de comportements suicidaires avec les ISRS (pour revue : http://www.nimh.nih.gov/health/topics/child-and-adolescent-mental-health/antidepressant-medications-for-children-and-adolescents-information-for-parents-and-caregivers.shtml).

En conclusion, les études mentionnées précédemment ont montré que les ISRS pourraient être intéressants dans le traitement des troubles paraphiles. Les ISRS sont probablement plus efficaces dans le traitement des troubles paraphiles qui ressemblent ou sont accompagnés par des symptômes de type obsessionnels ou dépressifs. Les indications recommandées pour l'utilisation des ISRS concernent principalement le traitement des troubles paraphiles mineurs ou des patients présentant des comorbidités souffrant de dépression ou de trouble obsessionnel-compulsif (Thibaut et al 2010 ; Bradford, 1999, 2000 ; Bradford et Federoff, 2006, 2013). Des recherches supplémentaires démontrant l'efficacité des ISRS dans le traitement des troubles paraphiles sont encore nécessaires et les études à long terme font défaut. Leur utilisation dans cette indication se fait jusqu'qu'alors hors AMM.

# Traitements antiandrogènes

Malgré l'efficacité des oestrogènes, des effets indésirables nombreux et graves ont été rapportés avec ces derniers (nausées, prise de poids, féminisation, cancer du sein, effets cardio-vasculaires et maladie ischémique cérébrovasculaire, thromboembolie) excluant leur utilisation chez les délinquants sexuels ou chez les sujets souffrant de troubles paraphiles. Même si de nombreuses études ont rapporté l'efficacité du traitement des délinquants sexuels avec l'acétate de médroxyprogestérone (MPA), le rapport bénéfice / risque semble ne pas favoriser l'utilisation du MPA, qui a été abandonné en Europe. En France, seule l'acétate de cyprotérone et les agonistes de la gonadolibérine sont utilisés dans cette indication.

# L'acétate de cyprotérone (CPA)

# Efficacité:

Le CPA (Androcur®) est un stéroïde synthétique, semblable à la progestérone, qui a une action progestative et antiandrogène. Le CPA agit par l'intermédiaire de sa liaison à tous les types de récepteurs aux androgènes, y compris les récepteurs du cerveau, bloquant l'absorption intracellulaire de la testostérone et son métabolisme. En effet, le CPA est un inhibiteur compétitif de la liaison de la testostérone et de la dihydrotestostérone (DHT) à des sites récepteurs androgènes. En outre, le CPA a une forte action progestative provoquant l'inhibition de la sécrétion de GnRH et une diminution à la fois de la GnRH et de la libération de LH (Jeffcoate et al 1980; Neuman, 1977). Le CPA est déjà enregistré dans plus de 20 pays dont la France pour la modération de la libido chez les hommes adultes atteints de déviations sexuelles ainsi que pour le cancer de la prostate non opérable (Androcur®) et il est principalement utilisé au Canada, au Moyen-Orient et en Europe (Thibaut et al, 2010). Le CPA peut être prescrit par voie orale sous forme de comprimés de 50 et 100 mg (50-200 mg / jour). L'utilisation clinique du CPA chez les



délinquants sexuels, principalement des exhibitionnistes, a été décrite pour la première fois en Allemagne (Laschet et Laschet, 1967 et 1971), dans une étude ouverte. Neuf rapports de cas, dix études en cross over sans comparatif en ouvert et double ou simple aveugle et enfin deux études comparatives en cross over et en double aveugle concernant le traitement de plus de 900 sujets de sexe masculin au total ont été rapportées dans la littérature. Une étude croisée en double insu comparant CPA et éthinyl-estradiol a conclu que les deux traitements avaient également diminué l'intérêt sexuel, l'activité sexuelle, sans effets indésirables majeurs (Bancroft et al., 1974). Une autre étude comparant le CPA et le MPA chez 7 délinquants sexuels a rapporté une efficacité équivalente sans effets indésirables, sauf ceux liés à hypoandrogénie (aucune analyse statistique n'a été effectuée) (Cooper et al., 1992). Parmi les études en double aveugle, une seule étude comparant CPA versus placebo et CPA versus absence de traitement, a effectué une analyse statistique et fait état d'une diminution statistiquement significative de l'activité sexuelle déviante (Bradford et Pawlak, 1993). Cinq autres études ouvertes ont rapporté l'utilisation du CPA (Laschet et Laschet, 1971; Laschet et Laschet, 1975; Bradford et Pawlak, 1993; Laschet et Laschet, 1971). Dans la plupart des études, le CPA est prescrit de 50 à 300 mg / jour per os ou par voie intramusculaire, 300-600 mg, tous les 1 ou 2 semaines. Sur une durée de 4 à 12 semaines, le CPA a entraîné une diminution significative des fantasmes sexuels, de l'activité et de la fréquence de la masturbation et, dans environ 80-90% des cas, une disparition complète du comportement sexuel déviant. En outre, les érections matinales, l'éjaculation et la spermatogenèse ont diminué. Ces auteurs ont suggéré que le CPA pourrait être utilisé, d'une manière dépendante de la dose, soit comme un agent de castration chimique soit comme un réducteur du désir sexuel, ce qui permet un maintien des capacités érectiles dans le cadre d'un comportement sexuel non déviant. L'efficacité a été maintenue alors que les patients étaient sous traitement pour une durée maximale de 8 ans dans un échantillon de 300 hommes souffrant de troubles paraphiles (CPA 50-200 mg/ jour par voie orale ou i.m. de 300-600 mg toutes les 1 ou 2 semaines) (Laschet et Laschet, 1975). Les effets du CPA sur l'activité sexuelle étaient totalement réversibles, un à deux mois après l'arrêt du traitement. L'efficacité du CPA chez cinq jeunes hommes ayant un comportement sexuel déviant ou une hypersexualité a été rapportée, cependant, le CPA ne devrait pas être prescrit avant la puberté car il a une incidence sur la croissance osseuse (Davies, 1974). Les taux de récidive ont été évalués dans sept études concernant un total de 127 personnes qui prennent du CPA (Meyer et Cole, 1997). Beaucoup de récidives ont été commises par des individus, qui n'avaient pas une bonne observance. À la fin du suivi (période de 2 mois à 4,5 ans), le taux moyen de récidive était de 6%. Il était environ 10 fois plus faible que le taux de 85% décrit avant le traitement.

Les concentrations sériques de FSH et de LH étaient soit diminuées soit inchangées par l'administration du CPA. Les taux de testostérone plasmatique étaient modérément diminués (Guay, 2009) et ne peuvent pas être utilisés comme marqueurs de l'observance du traitement.

# Effets indésirables liés à l'hypoandrogénie :

Asthénie, troubles du sommeil, symptômes ou troubles dépressifs, bouffées de chaleur, changements de pilosité, diminution du taux d'excrétion du sébum, crampes dans les jambes, chute de cheveux, réduction de la spermatogenèse (réversible), lmpuissance, diminution de l'activité sexuelle et des fantasmes, réduction du volume de l'éjaculat et ostéoporose (une fracture de hanche due à la perte minérale osseuse a été observée après 10 ans de traitement).

#### Effets indésirables liés au CPA:

Maux de tête, dyspnée, prise de poids, gynécomastie (20% des cas, réversible dans la plupart des cas), phénomènes thrombo-emboliques, augmentation du taux de prolactine, insuffisance surrénale ou hyperplasie (0,5% des cas chez les jeunes), hypertension artérielle, insuffisance



cardiaque, diminution de la tolérance au glucose, dysfonctionnement rénal, dysfonctionnement de l'hypophyse, anémie, douleurs locales au site d'injection (formulation retard), nausées, lésions hépatocellulaires (mais l'hépatotoxicité grave est rare ; observée dans moins de 1% des cas). Des antécédents thromboemboliques veineux ou une chirurgie récente augmentent le risque thromboembolique de 4 à 13 fois.

En conclusion, bien que de nombreuses études aient été publiées avec le CPA, la plupart des études ne sont pas contrôlées, et certains biais ont été observés (par exemple, la petite taille des échantillons, la courte durée de suivi dans la plupart des cas, les études ont été réalisées en crossover, la plupart sont des études rétrospectives). En outre, certains effets indésirables graves ont été observés avec le CPA et, dans certains pays, seule la forme orale est disponible et l'observance du traitement peut alors être erratique. Le taux de testostérone n'est pas systématiquement diminué et les mesures des concentrations plasmatiques du CPA ne sont pas disponibles dans de nombreux pays.

La dépendance hormonale du méningiome cérébral est bien connue, mais le CPA (acétate de cyprotérone) semble avoir une influence plus forte sur la croissance tumorale. Plusieurs études épidémiologiques récentes ont montré un risque accru de méningiome chez les personnes ayant reçu de fortes doses de CPA pendant au moins 6 mois (taux d'incidence de 60 pour 100 000 annéespersonnes contre 7 chez les non-utilisateurs (Gil et al., 2011). Chez les patients atteints de méningiome, le risque associé à une forte dose de CPA (OR 6,3 IC : 1,37-28,92) chez les hommes (3/745 patients utilisant actuellement une CPA) était nettement supérieur à celui observé chez les non-utilisateurs (Cea-Soriano et al., 2012). Dans 12/12 cas, une stabilisation de la croissance et une régression ont été rapportées après l'arrêt du traitement par le CPA sans reprise de croissance au cours d'une période de suivi moyenne d'un an (Bernat et al., 2015). En France, une IRM structurelle est recommandée par l'ANSM depuis juin 2019 avant le traitement en cas de traitement prolongé prévu (> 6 mois avec une dose élevée> 100 mg / jour). Ensuite, l'IRM doit être contrôlée à la 5e année, puis tous les 2 ans si le CPA est maintenu. Lorsque le CPA est arrêté, aucun suivi supplémentaire n'est requis. De rares cas de prolactinomes ou de somatotrophinomes ont été rapportés chez des transsexuels recevant des œstrogènes en association avec la CPA (Garcia-Malpartida et al. 2010 ; Nota et al., 2018). Cependant, le dépistage régulier des taux de prolactine n'est pas recommandé par ces auteurs.

#### • Les analogues de la gonadolibérine (GnRH)

Les analogues de la GnRH (GnRHa) sont en fait des agonistes de la GnRH qui agissent sur les récepteurs hypophysaires de la GnRH. Une augmentation transitoire de la testostérone, au début du traitement par les GnRHa est causée par une augmentation transitoire de la libération de LH, un phénomène appelé « flare-up ». Après cette stimulation initiale, l'administration continue des GnRHa permet d'obtenir une désensibilisation rapide des récepteurs de la GnRH et entraîne une réduction de la LH (et dans une moindre mesure de l'hormone folliculo-stimulante (FSH)) et ainsi de la testostérone à des niveaux équivalents à ceux obtenus avec une castration chirurgicale dans un délai de 2 à 4 semaines. Les GnRHa n'interférent pas avec l'action des androgènes d'origine surrénalienne. En outre, des neurones contenant de la GnRH envoient des projections dans l'hypophyse et dans des sites extra-hypophysaires, tels que le bulbe olfactif ou l'amygdale. Dans ces régions, les GnRHa peuvent avoir un effet neuromodulateur sur le comportement sexuel.

Trois analogues de la gonadolibérine (GnRH) sont disponibles: la triptoréline est un décapeptide de synthèse développé en tant que sel de pamoate (3 mg, formulation 1 mois ou 11,25 mg, formulation 3 mois), récemment approuvé en Europe pour la diminution réversible de la testostérone plasmatique à des niveaux de castration afin de réduire les pulsions sexuelles



déviantes des hommes adultes (triptoréline longue Durée d'Action 11,25 mg); La leuproréline a été développée sous forme intra musculaire d'administration quotidienne, ou sous forme retard avec des injections mensuelles (3,75, ou 7,5 mg, formulation 1 mois ou encore 11,25 mg, formulation 3 mois), ce dernier n'a pas d'AMM dans les troubles paraphiles; La goséréline a été développée sous forme injectable d'administration quotidienne, ou sous forme retard avec des injections mensuelles (3,6 ou formulation 1 mois 10,8 mg en sous-cutanée), et n'a pas d'AMM dans les troubles paraphiles. Peu d'études de cas (6 cas) ont rapporté l'efficacité de la goséréline, qui n'est pas utilisée dans cette indication en France.

En ce qui concerne le traitement des patients souffrant de troubles paraphiles, plusieurs études de cas et des études en ouvert ont été publiées. À ce jour, aucune étude randomisée n'a été publiée. Dans la plupart des études, le CPA ou le flutamide ont été simultanément utilisés pendant les premières semaines de traitement avec les GnRHa pour prévenir les conséquences d'un effet de « flare-up » sur le comportement sexuel. Dans la plupart des cas, une psychothérapie concurrente a été utilisée conjointement.

# Efficacité de la triptoréline

L'utilisation de la triptoréline a été décrite dans deux études ouvertes prospectives (41 hommes) (Rösler et Witztum, 1998; Thibaut et al 1993; Thibaut et al 1996; Thibaut et al 1998), une étude rétrospective (30 hommes) (Hansen et Lykke-Olesen, 1997) et une étude ouverte comparant différents GnRHa, y compris la triptoréline chez 3 sujets par rapport au CPA (Czerny et al, 2002). La majorité des patients traités par triptoréline pendant des durées de quelques mois à 7 ans (3,75 mg / mois) avaient soit une pédophilie soit un exhibitionnisme. Dans l'étude de Thibaut et al. (1993), le CPA a été utilisé pendant les premières semaines de traitement avec la triptoréline, afin d'éviter les conséquences sur le comportement d'un effet de « flare-up ». Dans toutes ces études, pendant la durée du traitement avec les GnRHa, aucun comportement sexuel déviant n'a été observé et aucune infraction sexuelle n'a été commise, sauf dans un cas. Parallèlement à une diminution rapide et forte de la testostérone et de la LH, une réduction des fantasmes et des comportements sexuels déviants et non déviants a été observée avec un effet maximal après 1 à 3 mois de traitement. Un tiers des cas (13 cas) avaient préalablement reçu du CPA seul sans efficacité. Après l'arrêt brutal du traitement dans 10 cas, (dans trois cas du fait d'effets indésirables liés aux GnRHa), le comportement et les fantasmes sexuels déviants sont réapparus dans sept cas sur 10. Dans trois cas, la triptoréline a été reprise avec une bonne efficacité et dans trois cas, le CPA (200 mg / jour) a été introduit, mais sans efficacité dans deux des trois cas. Dans un autre cas, la triptoréline a progressivement été interrompue en s'aidant de la supplémentation en testostérone chez un patient avec une perte minérale osseuse et aucune récidive n'a été observée. Dans une étude rétrospective, dans cinq cas, les sujets ont interrompu les GnRHa à leur sortie de prison, une rechute a été observée (Hansen et Lykke-Olesen, 1997).

# Efficacité de la leuproréline :

L'utilisation de la leuproréline a été décrite dans le traitement de 45 patients ayant des comportements paraphiles dans quatre études : trois études ouvertes et une étude rétrospective comparant la leuproréline et le CPA (Czerny et al 2002 ; Briken et al 2001 ; Briken 2002 ; Krueger et Kaplan, 2001 ; Schober et al 2005 ; Schober et al 2006). Le CPA ou le flutamide ont été utilisés en association avec les GnRHa au cours des premières semaines de traitement. Dans les quatre études, les troubles paraphiles les plus fréquemment observés étaient la pédophilie, le sadisme sexuel et l'exhibitionnisme. Des infractions sexuelles antérieures avaient été signalées dans 16 cas. La durée maximale du suivi était de 57 mois (durée moyenne environ 1 an). Schober et al. (2005) ont comparé la thérapie comportementale avec de l'acétate de leuprolide ou un placebo dans une



étude croisée chez cinq pédophiles. Dans trois cas, alors que les sujets recevaient un traitement placebo, les fantasmes sexuels déviants sont revenus et les niveaux de testostérone sont revenus aux niveaux de base. Dans une étude de cas (Briken et al., 2004), le patient a rechuté pendant le traitement par la leuproréline et a commis une infraction sexuelle.

Le CPA et les GnRHa ont montré la même efficacité incluant une absence d'effet sur le comportement sexuel déviant dans trois cas au sein de chaque groupe (58 sujets au total); une augmentation des fantasmes sexuels a même été signalée dans un cas avec un traitement par le CPA (Czerny et al., 2002). Dans deux cas précédemment traités avec le CPA, l'intensité du désir sexuel et des symptômes a été notablement réduite avec des GnRHa par rapport à un traitement antérieur par le CPA. La durée minimale de traitement nécessaire pour atteindre la disparition du comportement sexuel déviant et les conditions de l'arrêt du traitement restent en suspens. L'efficacité a été maintenue aussi longtemps que le traitement anti-androgène a été utilisé et la durée maximale de suivi a été de 7 ans pour la triptoréline et de 10 ans pour l'acétate de leuprolide. Dans l'étude de Rousseau et al. (1990), les auteurs ont rapporté une récidive lorsque le traitement avec la leuproréline et la flutamide a été brusquement arrêté à 26 semaines alors qu'il était efficace. Dans l'étude de Thibaut et al. (1996), les auteurs ont décrit la récurrence des comportements ou des fantasmes sexuels déviants dans les 8-10 semaines après interruption du traitement dans deux cas après, respectivement, 12 et 34 mois de traitement efficace avec les GnRHa. Dans ce dernier cas, le traitement GnRHa a été réintroduit et les fantasmes déviants ont de nouveau disparu. Dans un troisième cas, après 4,5 années de traitement efficace par les GnRHA, la testostérone a été progressivement ajoutée en raison d'une déminéralisation osseuse. Lorsque les GnRHa et la testostérone ont été arrêtés après 10 mois de prescription concomitante (dès que le niveau de testostérone était de retour à la normale), le comportement sexuel déviant n'est pas réapparu et l'absence de fantasmes ou de comportements sexuels déviants a duré jusqu'à 1 an après interruption du traitement. Dans l'étude de Rösler (1998), dans huit cas, la triptoréline a été interrompue après 8-10 mois et les troubles paraphiles ont repris dans cinq cas. Dans une étude rétrospective de Hansen (1997), cinq sujets ont arrêté la triptoréline quand ils ont quitté la prison et dans un cas, le comportement sexuel déviant est réapparu. Dans des études de cas supplémentaires, le comportement sexuel déviant a repris lorsque la triptoréline a été arrêtée en raison d'une déminéralisation osseuse (Hoogeveen et Van der Ver, 2008). Dans l'étude de Krueger et Kaplan (2001), dans un cas, l'acétate de leuprolide a été arrêté et un comportement sexuel déviant a réapparu. Dans l'étude de Schober (2005), où l'acétate de leuprolide a été remplacé par un placebo, dans trois des cinq cas, le comportement sexuel déviant est réapparu dans les 2 mois qui ont suivi l'arrêt et, dans un cas, il y avait un risque élevé d'infraction sexuelle. Selon l'expérience des différents auteurs, une durée minimale de 3 ans est nécessaire afin d'établir une relation stable avec le patient et de lui permettre d'accepter sa maladie et de la nécessité d'un traitement pharmacologique.

#### Effets indésirables GnRHa:

La perte minérale osseuse devrait être évaluée régulièrement chez les patients recevant un traitement par GnRHa. L'étude de Thibaut et al. (1996) (6 cas), a rapporté une diminution des valeurs de densité osseuse vertébrale et fémorale sans signes cliniques, mais nécessitant un suivi médical, au cours de la troisième année de traitement par la triptoréline chez un patient âgé de 27 ans. Dans l'étude de Rösler et Witztum (1998), l'effet de la triptoréline sur la densité minérale osseuse a été évalué chez 18 hommes par ostéodensitométrie avec un suivi séquentiel. Parmi ceux-ci, la densité minérale osseuse vertébrale ou fémorale a été réduite chez 11 hommes et inchangée chez les 7 autres. Deux patients présentant une déminéralisation osseuse progressive ont reçu des suppléments de calcium et de vitamine D par voie orale après 24 mois de traitement par la



triptoréline. Cinq autres cas de déminéralisation osseuse ont été observés dans des études de cas. Czerny et al. (2002) ont rapporté 1/29 cas de perte minérale osseuse avec des GnRHa. Grasswick et Bradford (2003) ont concentré leur étude sur la densité osseuse et rapporté une déminéralisation dans 2/4 des cas avec le CPA, un cas avec la leuproréline et dans 2/2 cas avec la castration chirurgicale. Les patients traités par GnRHa peuvent également présenter des bouffées de chaleur, une asthénie, des nausées, une prise de poids (2-13%), une douleur passagère ou une réaction cutanée au site d'injection, une diminution de la croissance des poils du visage et du corps (2-23%), des variations de la pression artérielle, une diminution de la tolérance au glucose, une diminution du volume des testicules (4-20%), une éjaculation douloureuse épisodique, une rigidité musculaire diffuse, une transpiration excessive, des symptômes dépressifs et une gynécomastie légère (2-7%).

En conclusion, même si aucune étude contrôlée n'a été réalisée et si certains biais ont été observés (petite taille des échantillons, courtes durées de suivi, conception des études ouvertes ou rétrospectives, hétérogénéité des sujets inclus), l'efficacité des GnRHa observée dans ces études en ouvert était très élevée. Il convient de souligner que, dans la plupart des cas décrits, les sujets avaient déjà été traités avec la psychothérapie, les ISRS ou d'autres anti-androgènes sans efficacité. En fait, en dépit de leur efficacité, les traitements par le MPA et le CPA sont associés à un pourcentage élevé d'effets indésirables qui limite considérablement leur utilisation, en particulier pour le MPA en Europe. En outre, une mauvaise observance du traitement est fréquemment observée avec le traitement par CPA sous forme orale. En revanche, les GnRHa sont plus puissants que le CPA ou le MPA. En outre, ils induisent moins d'effets indésirables, à l'exception de ceux relatifs à l'hypoandrogénie (Czerny et al., 2002). Les GnRHa peuvent être administrés par voie parentérale, une fois tous les un à trois mois, ce qui augmente l'observance du traitement. Les GnRHa devraient être utilisés quand d'autres solutions ont été écartées ou quand il y a un risque élevé de violence sexuelle. Les GnRHa constituent probablement le traitement le plus prometteur pour les délinquants sexuels à risque élevé de violence sexuelle, comme les pédophiles, les sadiques sexuels ou les violeurs en série.

# 2.3.3 Recommandations actuelles sur le traitement des paraphilies

En France (ainsi que dans de nombreux pays en Europe), dans un contexte de faibles preuves scientifiques, l'Agence française du médicament a approuvé deux traitements antiandrogènes chez les sujets paraphiles : l'acétate de cyprotérone a été approuvé pour la «modération du désir sexuel chez les hommes adultes atteints de déviance sexuelle" (Androcur® 100mg en comprimés); la triptoréline (Salvacyl®, 11,25 mg formulation à longue durée d'action par voie intramusculaire) a été approuvé dans l'indication "diminution réversible des taux de testostérone jusqu'à des niveaux de castration afin de diminuer le désir sexuel chez les hommes adultes atteints de déviance sexuelle".

Les ISRS ne sont pas encore approuvés dans le traitement des troubles paraphiles mais sont très souvent utilisés "hors AMM" sans preuves scientifiques en faveur de leur efficacité.

La "Haute Autorité de Santé" a publié des recommandations (2010) afin d'aider les cliniciens impliqués dans le suivi des agresseurs d'enfants (Recommandations nationales pour la prise en charge des auteurs d'agression sexuelle à l'encontre des mineurs de moins de 15 ans (Haute Autorité de Santé 2010 (<a href="http://www.has-sante.fr/portail/upload/docs/application/pdf/2010-03/aas-recommandations.pdf">http://www.has-sante.fr/portail/upload/docs/application/pdf/2010-03/aas-recommandations.pdf</a>). La fédération mondiale des sociétés de psychiatrie biologique (WFSBP) (F. Thibaut et al, World J Biol Psychiatry, WFSBP 2010;

(http://www.wfsbp.org/fileadmin/user\_upload/Treatment\_Guidelines/Paraphilias\_Guidelines.pdf

Florence Thibaut, Paul Cosyns, John Paul Fedoroff, Peer Briken, Kris Goethals, John M.



W. Bradford & The WFSBP Task Force on Paraphilias (2020) The World Federation of Societies of Biological Psychiatry (WFSBP) 2020 guidelines for the pharmacological treatment of paraphilic disorders, The World Journal of Biological Psychiatry, 21:6, 412-490, DOI:) a également publié des recommandations internationales concernant le traitement pharmacologique des paraphilies. Enfin, le ministère français de la Santé veut augmenter le niveau de connaissance sur l'utilisation de traitements pharmacologiques dans ces populations particulières de délinquants sexuels paraphiles (en termes d'efficacité et de tolérance).

Un algorithme (recommandations HAS et WFSBP) distingue six niveaux de traitement pour différentes catégories de paraphilies :

La psychothérapie est utilisée chez tous les délinquants (dans la plupart des cas, la thérapie comportementale est préférable). Chez les sujets paraphiles à risque élevé de récidive, le traitement pharmacologique devrait être utilisé comme traitement de première intention. La combinaison d'une psychothérapie et d'une thérapie pharmacologique est associée à une meilleure efficacité par rapport à un seul des deux traitements en monothérapie (Hall et Hall, 2007). Chaque niveau de traitement dépendra de la sévérité de l'affection paraphilique. Les traitements pharmacologiques (ISRS ou traitement anti-androgène) sont recommandés à partir du niveau 2.

#### **NIVEAU 1**

- Objectif : contrôle des fantasmes, pulsions et comportements sexuels paraphiles sans impact sur l'activité sexuelle conventionnelle et sur le désir sexuel
- Psychothérapie (thérapie comportementale et cognitive préférentiellement si disponible (niveau C), aucun niveau de preuve pour d'autres formes de psychothérapie

#### **NIVEAU 2**

- Objectif : contrôle des fantasmes, pulsions et comportements sexuels paraphiles avec un impact mineur sur l'activité sexuelle conventionnelle et sur le désir sexuel
- Peut être utilisé dans tous les cas bénins ("hands off" paraphiles à faible risque de violence sexuelle, à savoir l'exhibitionnisme sans risque de viol ou la pédophilie)
  - Pas de résultats satisfaisants au niveau 1
- ISRS : augmenter la dose au même niveau que dans les TOC (par exemple la fluoxétine à 40 à 60 mg/jour ou la paroxétine à 40 mg/jour (niveau C)

#### **NIVEAU 3**

- Objectif : contrôle des fantasmes, pulsions et comportements sexuels paraphiles avec une réduction modérée de l'activité sexuelle classique et du désir sexuel
  - paraphilies avec des caresses, mais sans pénétration
  - fantasmes sexuels paraphiles sans sadisme sexuel
  - Pas de résultats satisfaisants au niveau 2 après 4-6 semaines de ISRS à des doses élevées
- Ajouter un antiandrogène à faible dose (par exemple l'acétate de cyprotérone 50-100 mg / jour) à des ISRS (Niveau D)

# **NIVEAU 4**

- Objectif : contrôle des fantasmes, pulsions et comportements sexuels paraphiles avec une réduction substantielle de l'activité sexuelle et du désir
- Risque modéré élevé de violence sexuelle (paraphilie graves avec des caresses plus intrusives avec un nombre limité de victimes)
- Pas de fantasmes et / ou de comportement de sadisme sexuel (le cas échéant : passer au niveau 5)
  - bonne observance impérative, sinon : utilisation i.m. ou passer au niveau 5



- Pas de résultats satisfaisants au niveau 3
- Premier choix : pleine dose d'acétate de cyprotérone (CPA) : par voie orale, 200-300 mg / jour ou i.m. 200-400 mg une fois par semaine ou toutes les 2 semaines ; utiliser l'acétate de médroxyprogestérone : 50-300 mg/jour si le CPA n'est pas disponible (niveau C)
- En cas de comorbidité avec de l'anxiété, des symptômes dépressifs ou obsessionnels compulsifs, les ISRS peuvent être associés à l'acétate de cyprotérone

#### **NIVEAU 5**

- Objectif : contrôle des fantasmes, pulsions et comportements sexuels paraphiles avec une suppression quasi totale du désir et de l'activité sexuels
  - Risque élevé de violence sexuelle et paraphilies graves
  - fantasmes et/ou comportement de violence physique avec sadisme sexuel
  - Non-respect ou pas de résultats satisfaisants au niveau 4
- GnRHa, à savoir la triptoréline sous forme 3 mg/mois ou 11,25 mg i.m. tous les 3 mois (niveau C)
- Les niveaux de testostérone mesurés peuvent être facilement utilisés pour contrôler l'observance du traitement si nécessaire
- L'acétate de cyprotérone peut être associée à un traitement agoniste de la GnRH (une semaine avant et pendant le premier mois de traitement par les GnRHa) afin d'éviter un effet de « flare-up » et de contrôler le risque de rechute de comportement sexuel déviant associée à cet effet

#### **NIVEAU 6**

- Objectif : contrôle des fantasmes, pulsions et comportements sexuels paraphiles avec une suppression complète du désir et de l'activité sexuels.
  - Paraphilies les plus graves (cas catastrophiques)
  - Pas de résultats satisfaisants au niveau 5
- Utilisation de traitement anti-androgène, à savoir l'acétate de cyprotérone (50-200 mg/jour per os ou 200-400 mg une fois par semaine ou toutes les 2 semaines i.m.) ou l'acétate de médroxyprogestérone (300-500 mg/ semaine i.m. si le CPA n'est pas disponible) en plus des agonistes de la GnRH (Niveau D)
  - Les ISRS peuvent également être ajoutés (Absence de preuve)

#### 2.3.4 Conclusion

Notre étude sera très utile pour mieux définir la population d'hommes délinquants sexuels paraphiles et leur évolution selon la prise en charge au cours d'un suivi de 3 ans. Cette étude sera menée en conformité avec le protocole, les bonnes pratiques cliniques (BPC) et les exigences réglementaires applicables.

Une subvention précédente (PHRC 2010, Projet EPIPARA, code 2012/057 / HP) a eu pour but d'identifier les délinquants sexuels paraphiles recevant des traitements pharmacologiques en France. Environ 350 dossiers médicaux ont été identifiés dans 17 centres en France lors de l'étude précédente (environ 40 sujets recevaient des ISRS et 63 recevaient des traitements antiandrogènes (soit l'acétate de cyprotérone soit des agonistes de la GnRH)). Dans cette étude précédente, 345 hommes délinquants sexuels paraphiles (environ 2/3 de troubles pédophiles (l'inceste a été inclus dans cette catégorie qui représente environ un tiers des cas), avec une moyenne de 2 délits sexuels antérieurs, seulement 20% d'entre eux avaient des antécédents d'infractions non sexuelles) ont été identifiés. Les analyses préliminaires ont montré que près d'un tiers avaient déclaré des antécédents d'infraction sexuelle. Dans environ un tiers de la population, une dépendance à l'alcool et/ou aux drogues illicites a été observée. Un niveau d'éducation faible ou moyen a été décrit dans plus de 90% (<lycée). La plupart des sujets vivaient seuls (article soumis). Tous les



centres impliqués dans l'étude précédente sont prêts à participer à une étude de suivi naturalistique de 3 ans visant à évaluer l'efficacité et la tolérance des traitements pharmacologiques chez les délinquants sexuels.

Les recommandations actuelles de prescription des traitements pharmacologiques chez des sujets paraphiles préconisent soit les antidépresseurs sérotoninergiques soit les traitements antiandrogènes en plus du traitement psychologique (de préférence thérapie comportementale) selon le niveau de gravité du trouble paraphile et le risque de délinquance sexuelle (Recommandations de la Haute Autorité de Santé, 2010; Fédération mondiale des sociétés de psychiatrie biologique, Thibaut et al., 2010).

Jusqu'à présent, peu d'études menées sur des petites séries de patients ont été publiées et les connaissances scientifiques sur le traitement des délinquants sexuels paraphiles sont modestes (en particulier concernant les indications respectives des ISRS et des traitements antiandrogènes, l'efficacité et la tolérance de ces traitements).

En fait, nous allons utiliser une méthode de suivi naturaliste (durée : 3 ans) et nous concentrerons nos principaux objectifs sur deux questions principales qui sont importantes dans la pratique clinique et qui ont été soulevées par Khan et al. (Revue Cochrane 2015): (1) l'évolution des patients selon le type de prise en charge ; la tolérance des traitements qui sont habituellement utilisés pendant de nombreuses années chez des jeunes délinquants sexuels atteints de paraphilies sévères (population différente par rapport à des personnes âgées de cancer de la prostate).

Nous collecterons un échantillon salivaire (pour la génétique) conservé à température ambiante et deux échantillons sanguins stockés entre -20°C et -80°C afin de réaliser ultérieurement des études de génétique et d'épigénétique (le patient devra donner explicitement son consentement pour l'examen génétique).

# 2.4 DESCRPTION DES ACTES ET DES PROCEDURES AJOUTES PAR LA RECHERCHE

Nous collecterons un échantillon salivaire (pour la génétique) conservé à température ambiante et deux échantillons sanguins stockés entre -20°C et -80°C afin de réaliser ultérieurement des études de génétique et d'épigénétique dans le cadre d'éventuelles études futures (le patient devra donner explicitement son consentement pour l'examen génétique).

Nous évaluerons la densitométrie osseuse chez les patients recevant un traitement antidépresseur afin d'obtenir une population de référence en recevant pas d'antiandrogènes qui pourra servir de référence.

#### Limites

La plupart des chercheurs demandent aux participants d'évaluer leur excitation sexuelle en utilisant des échelles de type Likert comme dans notre étude. Aucune recherche sur les mesures de la fiabilité de la réponse subjective, comme la fiabilité test-retest, n'a été rapportée dans la littérature à ce jour. Fait intéressant, l'excitation sexuelle subjective et la perception de la réponse génitale sont fortement corrélées (Chivers et al., 2010).

La pléthysmographie pénienne (utilisant des stimuli érotiques audio ou visuels, pourrait être utilisée, mais, selon Marshall et Fernandez (2000), de nombreux biais méthodologiques peuvent limiter l'utilisation de cette technique, de sorte qu'elle ne sera pas utilisée dans cette étude. Surtout, cette technique n'est pas utilisée en Europe chez ce type de patients.

La rechute sera définie comme tout type d'infraction sexuelle, leur nombre sera évalué, mais devrait rester un événement rare (nombre attendu faible, risque d'infraction sexuelle estimée dans la littérature à environ 10-20% lorsque le traitement est régulièrement pris). Les rechutes seront analysées statistiquement si leur nombre est suffisant, mais ne peuvent pas être un objectif prioritaire en raison de leur rareté attendue.



L'évaluation du risque de rechute est un élément clé dans la prévention de la récidive chez les délinquants sexuels. Il est généralement admis que lors de l'évaluation du risque de récidive sexuelle, les évaluations actuarielles sont supérieures à un jugement clinique non structuré, mais l'évaluation du risque est encore mal connue (Hanson et Morton Bourgon 2009).

Les principaux coûts de ce projet sont les ressources humaines, qui sont coûteuses, y compris le coût de la collecte des données et le coût de la coordination de cette étude nationale qui comprend de nombreux centres dans différentes régions de France. Ce sera une grande quantité de travail supplémentaire pour signaler toutes ces données à l'aide d'un eCRF, qui n'a pas été précédemment utilisé en psychiatrie dans ces populations, une infirmière formée à cette recherche (utilisation de l'eCRF et passation des questionnaires) se déplacera au moins deux fois au cours de l'étude ainsi que le Dr Lamy (déplacement au cours de la période d'inclusion pour formation et éventuellement aide aux inclusions).

# 2.5 RESUME DES BENEFICES ET DES RISQUES PREVISIBLES ET CONNUS POUR LES PERSONNES SE PRETANT A LA RECHERCHE.

#### 2.5.1 Bénéfices attendus:

À notre connaissance, cette cohorte sera la plus grande population de délinquants sexuels paraphiles étudiés pendant la durée la plus longue à ce jour dans un champ où la recherche est insuffisante.

Ce vaste échantillon bénéficiant de soins de routine et suivis pendant 3 ans va nous permettre d'analyser l'évolution des patients selon la prise en charge reçue par leur psychiatre traitant.

En outre, cette analyse des pratiques cliniques sera cruciale pour améliorer nos connaissances sur les indications de ces traitements, qui pourraient éventuellement être revues en ce qui concerne leur efficacité et la tolérance, en particulier dans les cas les plus graves de délinquants sexuels avec paraphilie.

Une récente analyse Cochrane (Khan et al. 2015) a conclu que des recherches supplémentaires étaient nécessaires devant inclure des tailles d'échantillons plus grands sur de plus longues durées de suivi.

Un des avantages attendus par les victimes potentielles et les patients sera le suivant : si le rapport bénéfice / risque d'un traitement anti-androgène est acceptable, une formation médicale de tous les thérapeutes qui sont en charge des délinquants sexuels sera organisée afin d'améliorer leurs connaissances à propos de ces traitements (indications, efficacité, événements indésirables).

Parallèlement à l'éducation des enfants et au diagnostic, et à la prise en charge précoce des victimes de violence sexuelle, le traitement des délinquants sexuels est un élément clé dans la réduction de la violence sexuelle et de ses conséquences graves sur les victimes en particulier pour les délinquants sexuels les plus graves (sujets pédophiles et violeurs en série) (Gene et al, 2001; Thibaut F. Approche psychiatrique des Déviances Sexuelles Ed Springer Verlag, 2013; Hanson et al, 2014; Thibaut F. Abus Ed O Jacob 2015). Un rapport estime que l'abus sexuel des enfants a coûté 6.7 milliards d'euros en 2018-2019 au Royaume-Uni (seulement pour la prise en charge des victimes) (https://www.gov.uk/government/publications/the-economic-and-social-cost-of-contactchild-sexual-abuse/the-economic-and-social-cost-of-contact-child-sexual-abuse). Les conséquences personnelles et sociales des viols et violences sexuelles sont un problème majeur de santé publique (Felitti, 1991; Thibaut 2015); 90-95% des victimes ont des conséquences psychologiques et/ou (https://www.europeanceo.com/business-andphysiques rapport européen management/the-cost-of-sexual-assault/). Le coût annuel des violences sexuelles est estimé à 1.5 à



2% du produit intérieur brut soit environ 35 euros par habitant par an (<a href="https://www.europeanceo.com/business-and-management/the-cost-of-sexual-assault/">https://www.europeanceo.com/business-and-management/the-cost-of-sexual-assault/</a>).

#### 2.5.2 Risques attendus:

La systématisation du recueil d'événements et de la surveillance des effets des traitements ne constitue pas un risque supplémentaire par rapport à un suivi habituel. L'ostéodensitométrie fait partie des examens complémentaires envisagés lors d'un suivi classique, l'irradiation est très faible, moindre que pour une radiologie classique. Il n'y a pas de risque attendu avec les prélèvements. Les outils d'évaluation psychologique utilisés sont des outils cliniques classiques. Leur passation sera réalisée dans un contexte d'examen médical, ce qui permettra la reprise d'éléments émergents éventuels avec le praticien.

Au total, le risque peut être considéré comme minime.

# 3. OBJECTIFS DE LA RECHERCHE

# 3.1 OBJECTIF PRINCIPAL

Evaluation de l'évolution des symptômes sexuels chez les sujets paraphiles inclus dans l'étude (3 groupes de patients : patients sous antiandrogènes, patients sous ISRS et patients sans traitements pharmacologiques de type ISRS ou antiandrogène).

#### 3.2 OBJECTIFS SECONDAIRES

- 1. Estimation du taux de rechute (reprise d'un comportement sexuel déviant) et facteurs associés à la rechute. Les rechutes seront analysées statistiquement si leur nombre est suffisant, mais ne peuvent pas être un objectif prioritaire en raison de leur rareté attendue;
- 2. Le rôle des troubles psychiatriques concomitants, des troubles de la personnalité et de l'impulsivité dans l'efficacité du traitement, de l'observance (si traitement pharmacologique) et du risque de rechute sera étudié en tenant compte de la gravité et du type de troubles paraphiles ;
- 3. Déterminer les facteurs pouvant être associés à l'évolution des symptômes sexuels, à l'efficacité des traitements et aux effets indésirables potentiels ;
- 4. Analyse des éventuels effets indésirables chez les sujets sous traitements pharmacologiques (ISRS ou antiandrogènes versus sans traitements);
- 5. Les modifications des caractéristiques cliniques et cognitives des délinquants sexuels au fil du temps et leurs relations avec l'évolution des symptômes sexuels, l'observance (si traitement pharmacologique) et les risques de rechute seront analysées. En particulier, l'utilisation de pornographie, d'alcool et de drogues illicites, le rôle de l'hypersexualité comorbide et les caractéristiques cognitives telles que : les distorsions cognitives, l'empathie, le déni, seront étudiés dans cette population, en tenant compte de la gravité et du type de troubles paraphiles. La plupart de ces facteurs sont couramment acceptés comme prédicteurs valides de la réponse au traitement, malgré l'absence de recherche systématique pour soutenir ces hypothèses. Le déficit d'évaluation psychométrique pour mesurer ces facteurs contribue aux difficultés de la recherche dans ce domaine. Dans cette étude, nous allons utiliser des échelles d'évaluation spécifiques validées en français pour analyser l'hypersexualité et les caractéristiques cognitives connues pour être associées à la délinquance ;
- 6. Le rôle des trajectoires de vie, avec un focus particulier sur les antécédents de violence physique ou sexuelle et l'exposition à la pornographie durant l'enfance, dans l'efficacité du



- traitement dans les groupes traités, de l'observance et du risque de rechute sera étudié en tenant compte de la gravité et du type de troubles paraphiles ;
- 7. Estimation du nombre de sujets pour qui une modification de la prise en charge est proposée au cours de l'étude et analyse épidémiologique de ce groupe en termes de comorbidité, tolérance aux traitements, évolution des symptômes sexuels.

# 4. CONCEPTION DE LA RECHERCHE

#### 4.1 CRITERES D'EVALUATION DE LA RECHERCHE

# Critère d'évaluation principal

Évaluation du comportement sexuel paraphile en utilisant l'échelle d'évaluation de l'intensité du désir et des symptômes sexuels (ISDSS, échelle d'autoévaluation) à l'inclusion et tous les 3 mois (trois aspects du comportement sexuel seront évalués en précisant leur intensité et leur fréquence par semaine respectivement au cours du mois précédent: (1) l'intérêt et le désir, à l'aide d'une échelle allant de 0 (aucun) à 8 (maximum), (2) les pensées et les fantasmes, en utilisant une échelle allant de 0 (aucun) à 8 (maximum), et enfin (3) la mesure de l'activité sexuelle, la personne indique la nature et le nombre de l'activité sexuelle paraphile par semaine au cours du mois ayant précédé la visite (nombre de masturbations par semaine, nombre d'activités sexuelles de toute nature qui conduit à un orgasme). La moyenne des 3 scores sera utilisée (Rösler et Witztum, NEJM, 1998).

# Critères d'évaluation secondaires:

- 1. Les rechutes éventuelles seront évaluées lors des visites trimestrielles : qu'elles soient déclarées lors des entretiens ou connues par d'autres sources (notification par la famille, les soignants, la justice, etc....). Les rechutes seront enregistrées par l'investigateur et immédiatement signalée au coordinateur. En cas d'incarcération, le patient sortira de l'étude.
- 2. Diagnostic de troubles psychiatriques concomitants : critères DSM-5; évaluation des troubles de la personnalité : PDQ-4+ (à l'inclusion) ; Impulsivité : BIS 11 (à l'inclusion). Observance du traitement : pour tous les patients échelle abrégée Brief Adherence Rating Scale (BARS). Pour les patients traités à l'ISRS et aux antiandrogènes : la concentration plasmatique de la testostérone sera mesurée à l'inclusion et ensuite en cas de doute sur l'observance.
- 3. Facteurs génétiques (\*): prélèvement salivaire et prélèvement sanguin (le patient peut refuser ces prélèvements).
- 4. Analyse des éventuels effets secondaires signalés par le médecin en charge du patient ou par le patient lui-même : le type, la fréquence, le moment de survenue d'événements indésirables, ainsi que, le cas échéant, la nécessité d'une consultation médicale, d'une hospitalisation, d'un arrêt de travail, de modifications ou d'une interruption du traitement en raison d'effets indésirables, seront recueillis. Ceci nous permettra de comparer avec les groupes recevant des ISRS ou des antiandrogènes.
- 5. L'examen clinique à l'inclusion et tous les 3 mois :



- Gynécomastie cliniquement observable (présence ou absence), la mesure de la pression artérielle, du poids.
- Fonctionnement cognitif : échelle d'agression et de viol (MOLEST et RAPE scales) plus empathie et déni qui ont disparu par rapport au précédent écrit.
- Questionnaire AUDIT pour l'alcool (autoquestionnaire d'aide au repérage de la consommation excessive). La consommation d'alcool : (grammes d'alcool pur par jour, nombre maximal de verres par occasion et ancienneté de la consommation) (à l'inclusion et à M36).
- La Consommation de drogues illicites : type et quantité par jour, ancienneté de la consommation sera évaluée (à l'inclusion et tous les 3 mois).
- Hypersexualité : PATHOS / PEACCE pour le diagnostic ; Compulsive Sexual Behavior Inventory pour l'évaluation d'une hypersexualité si Pathos positive (≥ 3) (à l'inclusion et à M36). Evaluation du risque de violence sexuelle : STABLE 2007 et Static 99 (à l'inclusion et à M 36).
- Evaluation cognitive (MoCA) et Stroop (à l'inclusion et à M 36).
- 6. Evaluation des trajectoires de vie traumatiques : THQ Les trajectoires de vie traumatisantes seront évaluées à l'inclusion à l'aide de la version française du Questionnaire d'Histoire des Traumatismes (recherche de toutes sortes de traumatisme) (Trauma History Questionnaire (THQ)) (à l'inclusion).
- 7. Les modifications du plan de traitement seront vérifiées et notifiées lors des visites tous les trois mois

(\*) A l'inclusion, deux prélèvements pour la réalisation d'une étude génétique seront effectués ((le patient devra donner explicitement son consentement pour l'examen génétique). Un échantillon salivaire (1 pot plastique spécifique pour étude de génétique dans lequel le prélèvement salivaire sera réalisé, les échantillons salivaires se conservent à l'état ambiant. Ils seront rapatriés vers le centre INSERM U1266 par un transporteur spécialisé. Seront également prélevés deux tubes EDTA 4ml de sang (par un médecin ou une infirmière), ces tubes seront stockés entre -20°C et -80°C. Si un Centre de Ressources biologiques (CRB) est proche du lieu de prélèvement, les tubes sanguins seront stockés au CRB avant d'être acheminés à la fin de la première année d'inclusion vers le centre INSERM U1266 dans le laboratoire où travaille le Pr Thibaut. S'il n'y a pas de CRB proche du lieu de prélèvement, les tubes seront stockés dans un congélateur dédié à cet effet dans le centre d'inclusion. Un transporteur, à la fin des inclusions, sera chargé de faire parvenir l'ensemble des prélèvements au centre INSERM U1266.

Une collection biologique sera réalisée avec ces prélèvements.

#### 4.2 DESCRIPTION DE LA MÉTHODOLOGIE DE LA RECHERCHE

# 4.2.1 Plan expérimental

Le protocole de recherche adopte une approche observationnelle longitudinale dédiée à l'évaluation des résultats des différentes modalités de prise en charge pour les sujets présentant des troubles paraphiliques. L'étude est non randomisée et non comparative, mettant l'accent sur le suivi de trois groupes distincts: Groupe sous Traitement ISRS; Groupe sous Traitement Antiandrogène; Groupe sans Traitement Pharmacologique (intervention psychothérapeutique uniquement).



# Caractéristiques de l'Étude :

• Type d'Étude : Observationnelle de suivi

• Comparaisons : Non randomisée, non comparative

• Nombre de Groupes: 3

• **Multicentrique**: L'étude sera menée dans plusieurs centres de recherche afin d'assurer une représentation géographique étendue et une diversité des modalités de prise en charge.

Les principaux résultats de la recherche seront axés sur l'analyse des effets des différentes modalités de prise en charge. En particulier, l'étude vise à évaluer l'évolution des symptômes sexuels dans les groupes traités pharmacologiquement, estimer l'incidence des événements indésirables dans les groupes recevant un traitement ISRS ou antiandrogène, et analyser l'évolution symptomatique chez les sujets sans traitement pharmacologique. Cette approche permettra une évaluation approfondie des résultats cliniques liés aux différentes modalités de gestion des troubles paraphiliques.

Les prélèvements génétiques serviront à constituer une base de données permettant l'étude de facteurs de risque génétiques associés aux paraphilies.

#### Centres investigateurs:

Recherche multicentrique nationale

Nombre prévu de centres de recrutement : Voir la liste des centres.

# 4.3 DESCRIPTION DES MESURES PRISES POUR REDUIRE ET EVITER LES BIAIS

# 4.3.1 Biais de Sélection

L'étude sera séquentiellement proposée à tous les patients qui se présentent au centre expérimental et qui répondent aux critères d'inclusion et d'exclusion définis. Cette méthode garantit que chaque patient éligible ait la même chance de participer à l'étude, ce qui aide à obtenir un échantillon représentatif de la population cible. En veillant à une inclusion systématique de tous les patients éligibles, le risque de biais de sélection est réduit et la validité ainsi que la généralisation des résultats de l'étude sont renforcées.

#### 4.3.2 Identification des sujets

L'identification des sujets inclus dans la recherche fera l'objet d'une anonymisation systématique. Dans le cadre de cette recherche, les sujets seront identifiés de la façon suivante :

 $n^\circ$  centre (entre 1 et 4 positions numériques) –  $n^\circ$  ordre de sélection de la personne dans le centre (entre 1 et 4 positions numériques) - initiale nom - initiale prénom

Cette référence est unique et sera conservée pour toute la durée de la recherche.



# 5. DEROULEMENT DE LA RECHERCHE

| Personnes dont le | Qui informe et recueille | A quel moment la | A quel moment le |
|---|---|---|---|
| consentement est | le consentement de la | personne est | consentement de la |
| sollicité | personne | sonne informée | |
| La personne qui se<br>prête à la recherche | L'investigateur principal ou collaborateur médecin déclaré et formé à la recherche (médecin addictologue ou psychiatre) | en amont de | À l'inclusion |

Une fois inclus dans l'étude (après obtention du consentement éclairé), les délinquants sexuels paraphiles seront évalués au moment de l'inclusion dans l'étude par le médecin investigateur et par une infirmière formée et dédiée à l'étude, puis seront suivis pour évaluer les patients pendant 3 ans.

Il pourra être recruté plusieurs infirmières en fonction des besoins et des centres. Les sujets inclus seront tous suivis en consultation ambulatoire. Chaque psychiatre en charge des sujets inclus dans cette étude rendra compte des données cliniques, biologiques et épidémiologiques à l'inclusion et à intervalles réguliers, comme indiqué ci-dessous pendant 3 ans pour chaque patient (eCRF). L'infirmière ou les infirmières (recrutées pour ce projet) sera/ont formée(s) aux tests et questionnaires par le Pr Thibaut ou le Dr Lamy. L'infirmière pourra assurer conjointement le rôle de technicien de recherche, après formation, et aidera les psychiatres pour compléter les dossiers électroniques (sur site si nécessaire) et sera en charge de la vérification des fichiers et de la collecte de toutes les données manquantes. Elle s'assurera de la réalisation des prélèvements biologiques ainsi que de l'ECG. L'ECG sera interprété par le médecin du centre, le coordonnateur ou bien par un médecin cardiologue si le médecin du centre ne sait pas l'interpréter. La majorité des psychiatres impliqués dans le suivi de ces sujets ont leurs propres réunions nationales, 3 fois par an en en coordination étroite avec le Dr Lamy. Le Dr Lamy organisera une réunion par an avec les médecins investigateurs, y compris ceux n'appartenant pas à la Fédération. Les données qui seront recueillies par les enquêteurs, sont conformes aux directives nationales et internationales relatives à un suivi régulier des sujets paraphiles (Haute Autorité de Santé (HAS), et la Fédération mondiale des sociétés de psychiatrie biologique (WFSBP) et ne seront pas de nature à introduire des biais au cours du suivi, sauf pour l'ostéodensitométrie des patients sous ISRS et les prélèvements de l'étude de génétique.

#### 5.1 CALENDRIER DE LA RECHERCHE

- Durée de la période d'inclusion : 24 mois

Durée de participation de chaque patient : 3 ans

- Durée totale de la recherche : 5 ans

#### **5.2 VISITES**

# 5.2.1 Visite d'inclusion

Une fois les critères de sélection vérifiés (Diagnostic de paraphilie (critères DSM-5)) et l'information faite au patient, l'investigateur recueille son consentement éclairé daté et signé.



La visite d'inclusion (durée 4 à 5 heures) se poursuit par :

- Diagnostic de troubles psychiatriques concomitants à l'aide des critères DSM-5
- Évaluation des troubles de la personnalité à l'aide de l'échelle PDQ-4+
- Diagnostic d'hypersexualité (Echelle PATHOS / PEACCE utilisée pour diagnostiquer les sujets)
- AUDIT C et évaluation des consommations d'alcool et de drogues illicites
- Trajectoires de vie (THQ)
- Evaluation des fonctions cognitives par le MoCA et le Stroop (inhibition)
- Prélèvement salivaire et prélèvement sanguin (le patient peut refuser ces prélèvements)
- Echelles HAD et Beck pour évaluer l'anxiété, la dépression et les idées suicidaires éventuelles

Les questionnaires suivants seront utilisés au début et au cours du suivi à différents intervalles :

- Évaluation du comportement sexuel : Echelle d'évaluation de l'intensité du désir et des symptômes sexuels (ISDSS) (autoévaluation, comportement sexuel paraphile ou non paraphile),
- Traitements actuels et doses : une brève description du type de psychothérapie ou de la thérapie comportementale utilisée (technique, nombre et durée des séances par semaine), la date de début et la date de fin du traitement le cas échéant pour les patients sous traitement ISRS ou antiandrogènes
- Rapport de tout événement indésirable (par le patient et avec la CTCAE)
- BARS pour l'observance du traitement pour les patients sous traitement ISRS ou antiandrogènes
- Évaluation de la qualité de la vie (SF-36)
- Évaluation des symptômes anxieux, dépressifs et des idées suicidaires (BDI, BSSI, HAD)
- Evaluation du fonctionnement cognitif : Molest and Rape Scale, BES (empathie), échelle de Mc Kibben (déni et minimisation)
- Hypersexualité (CSBI)
- Impulsivité (BIS 11)
- Risque de violence sexuelle et non sexuelle, Static 99 et STABLE 2007
- Examen clinique et évaluation des consommations d'alcool et de drogues illicites (gynécomastie, glycémie à jeun, profil lipidique, NFS, fonctions hépatiques, fonctions rénales)
- L'évaluation de la qualité de vie (SF36)
- Mesures biologiques et mesure des niveaux de testostérone plasmatique et de la TeBG. Mesure du taux de prolactinémie à l'inclusion
  - Uniquement pour le groupe antiandrogènes ou ISRS
- ECG (fréquence cardiaque, recherche de troubles de la conduction cardiaque ou de troubles du rythme cardiaque) chez tous les patients traités (ISRS ou antiandrogènes) (RBP).
- Ostéodensitométrie (les Z scores des changements de densité osseuse vertébrale et fémorale seront analysés) (+/-7 jours)

Pour les patients qui ont donné leur consentement explicite, un prélèvement de salive et de sang sera effectué aux fins de l'étude génétique.

Toutes ces évaluations font partie de la surveillance de routine et ne doivent pas introduire de biais dans cette étude de suivi naturalistique de cohorte en dehors de l'ostéodensitométrie (dans le groupe ISRS). Les autres prélèvements font partie du bilan initial. Les variables



sociodémographiques et cliniques seront recueillies par le médecin investigateur, avec l'aide de l'infirmière si nécessaire : ces données sont généralement recueillies au cours des entretiens médicaux conformément aux recommandations nationales et internationales concernant la surveillance des sujets paraphiles (recommandations HAS et WFSBP) et n'introduiront pas de biais au cours du suivi (étude de soins de routine). Les antécédents personnels et familiaux de troubles psychiatriques ou de paraphilies et leurs traitements éventuels; les antécédents de traumatisme crânien avec PDC et l'âge de survenue; la notion de phymosis ou d'intervention sur les organes sexuels, l'âge d'exposition à la pornographie seront recueillis à l'inclusion ce qui est habituel en psychiatrie courante.

Durée totale de l'évaluation à l'inclusion : maximum 1 journée (si la durée d'évaluation dépasse 3h30, un repas ou une collation sera prévue pour le patient). Même si la plupart des échelles sont en auto-évaluation, l'infirmière formée aux évaluations devra recueillir les échelles d'auto-évaluation et avoir une brève discussion avec le sujet sur chaque échelle. Elle vérifiera qu'il n'y a pas de données manquantes dans les auto-évaluations.

L'infirmière (ou les infirmières) sera encadrée par le Pr Thibaut et le Dr Lamy et formée par ses soins aux échelles utilisées dans l'étude.

#### 5.2.2 Visites de suivi de la recherche

Les visites de suivi auront lieu tous les 3 mois (+/- 7 jours).

Le détail du déroulement des visites est précisé dans le « tableau récapitulatif de la chronologie de la recherche ».

Chaque visite durera environ 30 minutes.

- ISDSS (échelle d'évaluation de l'intensité du désir des symptômes sexuels) (autoquestionnaire)
  - Effets indésirables (rapportés par le patient et le CTCAE)
  - Poids, pression artérielle
  - Gynécomastie
  - Fonctions hépatiques (si l'acétate de cyprotérone est utilisé)
  - Rechute
  - BARS
  - Usage d'alcool et de drogues illicites
  - Traitements actuels et doses
  - Type de psychothérapie et fréquence
  - BDI-II, HAD
  - BSSI

#### 5.2.3 Visite de fin de la recherche

Seront réalisés (entre autres, cf tableau récapitulatif de la chronologie de la recherche) :

- L'évaluation de la qualité de vie (SF36), les échelles cognitives (Molest and Rape scale, BES, grille d'évaluation du déni et de la minimisation, BIS 11, CSBI si pathos ≥ 3 à l'inclusion, l'échelle de risque de récidive Static 99 et STABLE 2007.
- L'examen clinique cardiaque standard
- Les examens biologiques suivants : hépatique, rénal, glycémie à jeun, profil lipidique, NFS.



Uniquement pour le groupe antiandrogènes ou ISRS

- L'ostéodensitométrie (+/- 7 jours)
- L'ECG pour les patients traités.

# a. Tableau ou schéma récapitulatif de la chronologie de la recherche

| VISITES | Mois<br>M0<br>Inclusion | M3<br><u>+</u><br>1<br>sem | M6<br>±<br>1<br>sem | M9<br>±<br>1<br>sem | M12<br>±<br>1<br>sem | M15<br>±<br>1<br>sem | <u>+</u><br>1 | <u>+</u><br>1 | M24<br>±<br>1<br>sem | M27<br>±<br>1<br>sem | M30<br>±<br>1<br>sem | M33<br>±<br>1<br>sem | M36<br>Final |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Information et vérification des critères d'éligibilité | х | | | | | | | | | | | | |
| Consentement écrit | х | | | | | | | | | | | | |
| Données sociodémographiques | х | | | | | | | | | | | | |
| Antécédents (personnels, familiaux de troubles psychiatriques.) / médicamenteux | Х | | | | | | | | | | | | |
| Traitements actuels et doses Si traitement Type de psychothérapie et fréquence | х | х | х | х | х | х | Х | х | х | х | х | х | х |
| ISDSS (échelle d'évaluation de l'intensité du désir des symptômes sexuels) (autoquestionnaire) | х | х | х | х | х | х | х | х | х | х | х | х | х |
| Recherche d'une rechute : reprise d'un comportement sexuel déviant | x | х | х | х | х | X | х | х | X | х | х | х | x |
| Examen clinique (Poids et périmètre abdominal, taille, pression artérielle, recherche de gynécomastie) | х | х | х | х | х | X | х | х | х | х | х | х | х |
| Examen cardiaque | x | | | | | | | | | | | | Х |
| Recueil bilans biologiques (NFS,<br>Glycémie à jeun, profil lipidique,<br>fonctions rénales) | Х | | | | | | | | | | | | х |
| Fonctions hépatiques | x | * | * | | * | | * | | * | | * | | x |
| Taux testostérone plasmatique** avec TeBG et prolactinémie | х | | | | | | | | | | | | |
| Evénements indésirables (patient's report and CTCAE) | x | х | х | х | х | X | х | х | X | х | х | х | х |
| SF-36 short form | х | | | | | | | | | | | | х |
| Ostéo<br>Densitométrie (+/- 7 jours) * | x | | | | | | | | | | | | х |
| ECG (Si traitement) | Х | | | | | | | | | | | | Х |
| Prélèvement salivaire et prélèvement sanguin | х | | | | | | | | | | | | |
| BARS (observance) | х | х | Х | Х | х | Χ | X | Х | Х | Х | Х | Х | х |
| PDQ-4+ (troubles psychiatriques) | х | | | | | | | | | | | | |
| BIS 11 (impulsivité) | Х | | | | | | | | | | | | Х |


| VISITES | Mois<br>M0 | M3<br><u>+</u> | M6<br>+ | M9<br><u>+</u> | M12<br><u>+</u> | | | | M24<br><u>+</u> | M27 | M30<br><u>+</u> | M33<br>+ | M36 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Inclusion | 1<br>sem | ±<br>1<br>sem | 1<br>sem | 1<br>sem | <u>+</u><br>1<br>sem | 1<br>1<br>sem | ±<br>1<br>sem | 1<br>sem | ±<br>1<br>sem | 1<br>sem | ±<br>1<br>sem | Final |
| PATHOS/PEACCE (hypersexualité) | Х | | | | | • | | | · | | | | Х |
| CSBI (comportement sexuel compulsif) | X<br>Si PATHOS <u>≥</u> 3 | | | | | | | | | | | | X<br>Si<br>PATH<br>OS <u>&gt;</u><br>3 |
| Fonctionnement cognitif : BES (empathie) | х | | | | | | | | | | | | х |
| Fonctionnement cognitif: Molest and Rape Scale (distorsions cognitives) | x | | | | | | | | | | | | x |
| Fonctionnement cognitif: | | | | | | | | | | | | | |
| Grille d'Évaluation du Déni et de la<br>Minimisation | x | | | | | | | | | | | | x |
| Fonctionnement cognitif: | | | | | | | | | | | | | |
| Mo CA | х | | | | | | | | | | | | х |
| Stroop | х | | | | | | | | | | | | х |
| Static 99 | x | | | | | | | | | | | | Х |
| STABLE 2007 | Х | | | | | | | | | | | | Х |
| AUDIT C (conso excessive d'alcool) | Х | | | | | | | | | | | | Х |
| Utilisation d'alcool et de drogues | х | х | х | х | х | X | X | X | X | х | х | х | х |
| THQ (histoire des traumatismes) | х | | | | | | | | | | | | |
| BDI-II et HAD | x | х | | | x | | | | x | | | | x |
| BSSI | х | х | | | х | | | | х | | | | х |

<sup>\*</sup> seulement si antiandrogènes ou ISRS

#### Légendes

- PATHOS / PEACCE : Echelle pour le diagnostic d'hypersexualité
- PDQ-4+ : Personality Diagnostic Questionnaire version 4 (autoévaluation des troubles de personnalité)
- AUDIT C (dépistage d'un mésusage d'alcool recommandations HAS)
- Trajectoires de vie : THQ : Trauma Histoire questionnaire ;
- Fonctions cognitives (MoCA) et Stroop
- ISDSS : échelle d'évaluation de l'intensité du désir et des symptômes sexuels (auto évaluation)
- Les traitements actuels (type de médicaments, date de la première utilisation, et dose par jour) si un changement préciser le type et le dosage

Auto-évaluation de tout événement indésirable et CTC : Critères de terminologie commune pour les événements indésirables 4.0

<sup>\*\*</sup>en cours de traitement antiandrogène si l'acétate de cyprotérone est utilisé si doute sur observance



BARS : Brève adhésion Rating Scale (observance du traitement) - pour les patients sous traitement pharmacologique)

- SF-36 échelle : échelle pour évaluer la qualité de la vie dans sa forme courte (auto évaluation)
- BDI-II : Beck Depression Inventory (symptômes dépressifs)
- HAD Hospital Anxiey Depression Scale
- BSSI : Beck Échelle d'idéation suicidaire
- Evaluation du fonctionnement cognitif : Echelle de molestation et de viol (distorsions cognitives) (Molest and Rape Scale)
- Evaluation du fonctionnement cognitif : échelle d'empathie (BES)
- Evaluation du fonctionnement cognitif : grille d'évaluation du déni et de la minimisation de Mc Kibben
- Evaluation des fonctions cognitives (MoCA) et Stroop
- BIS 11 : échelle d'évaluation de l'impulsivité
- CSBI : échelle de mesure du comportement sexuel compulsif Hypersexualité
- Static 99 et STABLE 2007 : échelle d'évaluation du risque de violence sexuelle et non sexuelle
- Le profil lipidique comprend : le cholestérol total, les triglycérides, le cholestérol HDL
- La fonction hépatique comprend : ASAT, ALAT, bilirubine totale, gamma-glutamyl transférase et phosphatases alcalines.
- La fonction rénale comprend : urée sanguine et créatinine sérique.
- Numération formule sanguine.
- Mesures biologiques et mesure des niveaux de testostérone plasmatique systématique chez les délinquants sexuels pour éliminer une pathologie organique de l'axe gonadotrope TeBG: protéine transporteuse de la testostérone qui permet d'évaluer le taux de testostérone libre seule forme active qui n'avait pas été précisée mais est indispensable pour évaluer la testostérone libre seule forme active. Mesure à l'inclusion de la prolactinémie plasmatique (pour éliminer un prolactinome).
- Ostéodensitométrie (les Z scores des changements de densité osseuse vertébrale et fémorale seront analysés).
- ECG (fréquence cardiaque, recherche de troubles de la conduction cardiaque ou de troubles du rythme cardiaque).

## b. Distinction soin-recherche

Tableau : Distinction entre les actes liés au « soin » et les actes ajoutés par la « recherche »

| Interventions réalisées dans<br>le cadre de la recherche | Actes, procédures et traitements<br>liés aux <u>soins</u> | Actes, procédures ajoutées par <u>la recherche</u> |
|---|---|---|
| Consultations | Toutes les consultations sont<br>prévues dans le cadre des soins<br>courants | |
| Prises de sang | <ul> <li>Pour tous les sujets à l'inclusion et à M36 : glycémie à jeun, profil lipidique, NFS, fonctions hépatiques, fonctions rénales conformément aux BPC</li> <li>Pour les sujets sous</li> </ul> | donné leur consentement<br>explicite : tube de sang et |



| | antiandrogènes : fonctions<br>hépatiques à chaque consultation<br>conformément aux BPC | |
|---|---|---|
| Imagerie | Pour les sujets ayant un traitement pharmacologique type ISRS et antiandrogène à l'inclusion et à M36 : ECG à l'inclusion et M36 conformément aux BPC Pour les sujets sous antiandrogène : ostéodensitométrie à l'inclusion conformément aux BPC et à fin étude | Pour les sujets sous ISRS :<br>ostéodensitométrie à<br>l'inclusion et à la fin de<br>l'étude |
| Examen clinique | Poids et périmètre abdominal, examen cardiaque, pression artérielle, recherche de gynécomastie ISDSS, SF-36, recherche rechute, PDQ4+, BIS 11, PATHOS/PEACCE, CSBI si pathos ≥ 3, BES, Tests cognitifs (Grille d'évaluation du déni et | |
| Questionnaires<br>autoquestionnaires | minimilisation, MoCA), Static 99,<br>STABLE 2007; AUDIT C, THQ,<br>questionnaires pour évaluer les<br>traitements actuels, type de<br>psychothérapie et fréquences, BDI<br>II et HAD.<br>Pour les sujets sous<br>antiandrogènes et ISRS: BARS, | |

### c. Collection Biologique

Les échantillons issus des prélèvements sanguins et salivaires réalisés dans le cadre de la recherche feront l'objet de collections biologiques, en vue de recherches ultérieures. Ces échantillons ne feront pas l'objet d'analyses pendant la recherche.

Au cours de la recherche, ces échantillons destinés aux collections biologiques seront centralisés et conservés à l'institut de Psychiatrie et Neurosciences à Paris (unité INSERM U 1266) sous la responsabilité du Pr THIBAUT.

L'échantillon salivaire se conserve à température ambiante et les prélèvements sanguins (deux tubes EDTA 4ml de sang) sont stockés dans un congélateur (entre -20° et -80° C).

Les échantillons biologiques conservés pourront faire l'objet de recherche génétiques futures sur une meilleure compréhension des comportements à l'origine des délits sexuels. Ces échantillons pourront également être utilisés pour des analyses ultérieures non prévues dans le protocole pouvant se révéler intéressantes dans le cadre de la pathologie, en fonction de l'évolution des connaissances scientifiques, sous réserve que le patient n'y soit pas opposé, après en avoir été informé, comme indiqué dans le formulaire d'information/consentement de cette étude. Les prélèvements restants non utilisés lors des analyses seront systématiquement détruits.

A la fin de la recherche, ces collections biologiques seront déclarées auprès du ministère chargé de la recherche.



| Type de<br>prélèvement | Quantité | Lieu de conservation | Responsable<br>de la<br>collection | Finalité<br>de la<br>collection | Durée de la<br>conservation |
|---|---|---|---|---|---|
| Salive | 1 pot de salive | T° ambiante | Pr THIBAUT | Etude de<br>génétique | Collection biologique |
| Sanguin | 2 tubes<br>EDTA 4ml<br>de sang | Entre -20°C et -<br>80°C | Pr THIBAUT | Etude de<br>génétique | Collection<br>biologique |

#### 6. CRITERES D'ELIGIBILITE

#### **6.1 CRITERES D'INCLUSION**

- Hommes souffrant de paraphilies (critères DSM-5),
- Agés de 18 à 65 ans,
- Délinquants sexuels (délit ou agression à caractère sexuel incluant exhibitionnisme, viol, attouchement sexuel, inceste, détention de matériel vidéo à caractère pédopornographique) (niveau de gravité 1 à 6 selon les recommandations de la WFSBP),
- Sujet ayant donné son consentement,
- Patients pris en charge par la sécurité sociale,
- Maîtrise satisfaisante du français écrit et parlé.

#### **6.2 CRITERES DE NON INCLUSION**

- Sujet en prison (quel qu'en soit le motif),
- Sujet sous mesure de tutelle (les patients sous curatelle pourront en revanche être inclus),
- Les sujets ayant commis une infraction sexuelle et qui ne répondent pas aux critères DSM-5 de paraphilie,

#### **6.3 MODALITES DE RECRUTEMENT**

Le Dr Lamy est chargée d'être en contact avec les différents centres incluant des patients et de récupérer les CV des médecins investigateurs. L'infirmière, sous la coordination du Pr Thibaut, contactera les centres afin de préparer les inclusions des patients. L'objectif étant d'inclure l'ensemble des patients d'un même centre dans le même temps. Une journée de formation a déjà été réalisée afin que les investigateurs puissent se former aux passations des échelles de récidive (avec le Dr Ducro). Le reste de la formation de l'infirmière sera effectué par le Pr Thibaut.

Chaque sujet inclus recevra un numéro unique de code. Ce numéro sera utilisé lors de l'étude de suivi afin d'anonymiser de façon stricte chaque sujet inclus pendant toute l'étude. Ceci est notre préoccupation majeure dans cette population et nous allons accorder une attention particulière à la confidentialité à toutes les étapes comme nous l'avons fait lors de l'étude préliminaire nationale menée en vue d'identifier les délinquants sexuels paraphiles recevant des traitements pharmacologiques. Les sujets qui reçoivent déjà un ISRS ou des antiandrogènes ou aucun des deux au moment de l'inclusion seront inclus dans cette étude (le choix sera fait par les psychiatres traitants avec leurs patients). Nous n'interférerons pas avec le choix du type de prise en charge pour ne pas introduire de biais dans cette étude.



| Nombre total de sujets sélectionnés | 200 |
|-------------------------------------|-----|
| Période d'inclusion (mois) | 24 |
| Nombre des sujets / centre | 20 |

## 7. REGLES D'ARRÊT

Toute personne incluse dans la recherche peut quitter l'étude à tout moment et quelle qu'en soit la raison, en retirant son consentement. Les personnes dans ce cas seront sorties de l'étude.

## 7.1 CRITÉRES ET MODALITES D'ARRÊT PRÉMATURÉ DE LA RECHERCHE

Tout patient inclus dans la recherche peut à tout moment et quelle qu'en soit la raison retirer (ou le représentant légal) son consentement de participation. Dans ce cas, le patient sera sorti de l'étude.

L'investigateur peut interrompre temporairement ou définitivement la participation d'un patient à la recherche pour toute raison ayant un impact sur sa sécurité ou qui servirait au mieux les intérêts du patient. Dans tous les cas l'investigateur notera pour le patient considéré la date et les raisons de l'interruption prématurée.

En, cas d'arrêt prématuré de la participation du patient à la recherche ou de retrait de consentement, les données le concernant recueillies avant l'arrêt prématuré ou le retrait de consentement, pourront être utilisées, sauf si le patient ou le représentant légal, s'y oppose.

## 7.2 MODALITES DE REMPLACEMENT DE CES PERSONNES, LE CAS ÉCHÉANT

Les patients sortis prématurément de l'étude ne seront pas remplacés.

#### 7.3 ARRÊT D'UNE PARTIE OU DE LA TOTALITÉ DE LA RECHERCHE

Le promoteur GHU Paris ou le comité de protection des personnes (CPP) peuvent interrompre prématurément de façon temporaire ou définitive toute ou une partie de la recherche, dans les situations suivantes :

- des faits imprévus, de nouvelles informations relatives aux procédures, au vu desquels les objectifs de la recherche ou du programme clinique ne seront vraisemblablement pas atteints, peuvent amener le Promoteur ou l'Autorité Compétente (CPP) à interrompre prématurément la recherche,
- le Promoteur se réserve le droit de suspendre définitivement les inclusions, à tout moment, s'il s'avère que les objectifs d'inclusion ne sont pas atteints.

## 7.3.1 Modalités et calendrier de recueil pour ces données

En cas d'arrêt de la recherche ou du retrait du consentement, les données seront recueillies lors des visites prévues par le protocole et ce jusqu'au moment de l'arrêt de la recherche ou du retrait du consentement.



## 7.3.2 Modalité de suivi de ces personnes

En cas d'arrêt de la recherche ou du retrait du consentement les patients continueront à être suivis par leur psychiatre traitant conformément à la prise en charge habituelle.

## 8. VIGILANCE

Dans le cadre de cette étude, les événements indésirables (graves ou non) ne sont pas à notifier au promoteur. La notification doit se faire dans le cadre de la vigilance mise en place dans le cadre du soin pour la pratique faisant l'objet de la recherche.

## 8.1 COMITÉS SPÉCIFIQUE DE LA RECHERCHE

Il s'agit d'une étude observationnelle de suivi d'une cohorte de patients.

Le Pr Thibaut est le coordonnateur de l'étude.

Le Dr lamy et l'infirmière seront chargés de la coordination des différents sites. Les psychiatres traitants continueront à réaliser les soins courants de leurs patients. Il n'est pas prévu dans l'étude de comités spécifiques de la recherche.

#### 8.2 COMITÉ DE SURVEILLANCE INDÉPENDANT

Dans le cadre de cette étude à risques et contraintes minimes, il n'est pas jugé utile de nommer un CSI dans la mesure où aucun effet indésirable lié à l'étude n'est attendu et aucune surveillance particulière n'est à prévoir.

## 9. GESTION DES DONNÉES

## 9.1 MODALITÉ DE RECUEIL DES DONNÉES

Seules les données strictement nécessaires et pertinentes et prévues par le protocole au regard des objectifs de la recherche seront recueillies.

## 9.1.1 Accès aux données

#### Conformément aux BPC:

- le promoteur est chargé d'obtenir l'accord de l'ensemble des parties impliquées dans la recherche afin de garantir l'accès direct à tous les lieux de déroulement de la recherche, aux données source, aux documents source et aux rapports dans un but de contrôle de qualité et d'audit par le promoteur.
- les investigateurs mettront à disposition des personnes chargées du suivi, du contrôle de qualité, en cas d'audit de la recherche impliquant la personne humaine, les documents et données individuelles strictement nécessaires à ce contrôle, conformément aux dispositions législatives et réglementaires en vigueur.



#### 9.1.2 Accès aux documents source

Les documents source étant définis comme tout document ou objet original permettant de prouver l'existence ou l'exactitude d'une donnée ou d'un fait enregistré au cours de la recherche seront conservés pendant 15 ans par l'investigateur ou par l'hôpital s'il s'agit d'un dossier médical hospitalier.

Dans le cadre de cette recherche les documents source sont : le dossier médical, original de résultat d'examen biologique, compte-rendu d'examen d'imagerie, l'ECG

#### a. Confidentialité des données

Les personnes chargées du contrôle de qualité d'une recherche impliquant la personne humaine (article L.1121-3 du code de la santé publique), prendront toutes les précautions nécessaires en vue d'assurer la confidentialité des informations relatives à la recherche, aux personnes qui s'y prêtent et notamment en ce qui concerne leur identité ainsi qu'aux résultats obtenus.

Ces personnes, au même titre que les investigateurs eux-mêmes, sont soumises au secret professionnel (selon les conditions définies par les articles 226-13 et 226-14 du code pénal).

Pendant la recherche impliquant la personne humaine ou à son issue, les données recueillies sur les personnes qui s'y prêtent et transmises au promoteur par les investigateurs (ou tous autres intervenants spécialisés) seront rendues non identifiantes.

Elles ne doivent en aucun cas faire apparaître en clair les noms des personnes concernées ni leur adresse.

Seules les initiales du nom et du prénom seront enregistrées, accompagnées d'un numéro codé propre à la recherche indiquant l'ordre d'inclusion des sujets.

Le promoteur s'assurera que chaque personne qui se prête à la recherche a donné son accord par écrit pour l'accès aux données individuelles la concernant et strictement nécessaires au contrôle de qualité de la recherche.

# 9.2 TRAITEMENT DES DONNÉES ET CONSERVATION DES DOCUMENTS ET DES DONNÉES

# 9.2.1 Identification du responsable et du lieu de la gestion du traitement des données

La gestion du traitement des données et les analyses statistiques s'effectueront au sein de la DRCI du GHU Paris par la Cellule Biométrie.

## 9.2.2 Saisie des données

<u>eCRF</u> : La saisie des données rendues non identifiantes sera réalisée sur un support électronique via un navigateur internet.

L'analyse des données sera réalisée par nos soins. Les données seront saisies sur un eCRF (REDCap.



#### 9.2.3 Traitement des données (CNIL)

Cette recherche entre dans le cadre de la « Méthodologie de Référence pour les traitements de données personnelles opérés dans le cadre des recherches impliquant la personne humaine » (MR-001 Le GHU Paris, promoteur de la recherche, a signé un engagement de conformité à cette « Méthodologie de Référence »

Le traitement des données à caractère personnel de cette recherche est réalisé conformément au chapitre IX de la loi du 6 janvier 1978 relative à l'informatique, aux fichiers et aux libertés, modifiée (articles 53 à 61).

## 9.2.4 Archivage

Les documents spécifiques d'une recherche impliquant la personne humaine à risque et contraintes minimes seront archivés par l'investigateur et le promoteur pour une durée de 15 ans après la fin de la recherche.

Cet archivage indexé comporte notamment :

- Une enveloppe scellée pour l'investigateur contenant un exemplaire des formulaires de consentement signés de toutes les personnes du centre ayant participé à la recherche ;
- Une enveloppe scellée pour le promoteur contenant un exemplaire des formulaires de consentement signés de toutes les personnes du centre ayant participé à la recherche ;
- Les classeurs « recherche » pour l'Investigateur et le promoteur comprenant (liste non exhaustive) :
- Les versions successives du protocole (identifiées par le n° et la date de version), ses annexes
- Les avis du CPP
- Les courriers de correspondance,
- La liste ou registre d'inclusion,
- Les annexes spécifiques à la recherche
- Le rapport final de la recherche.
- Les documents de recueil des données.

### 9.3 PROPRIÉTÉS DES DONNÉES

Le Promoteur est propriétaire des données et aucune utilisation ou transmission à un tiers ne peut être effectuée sans son accord préalable.

## **10. ASPECTS STATISTIQUES**

### 10.1 DESCRIPTION DES MÉTHODES STATISTIQUES PRÉVUES

Étant donné leurs caractéristiques potentiellement différentes, les trois groupes (patients recevant des ISRS, patients recevant des antiandrogènes et patients ne recevant ni ISRS ni antiandrogènes) seront analysés séparément dans un premier temps. Si leurs caractéristiques à l'inclusion ne sont pas en contradiction avec l'hypothèse de positivité (probabilité de recevoir chacun des traitements conditionnelle aux caractéristiques non nulle et strictement inférieure à un), l'incidence d'effets indésirables et l'évolution de des symptômes sexuels pourront être comparées entre les trois groupes, ou entre deux groupes, après ajustement sur les différences à l'inclusion par pondération ou par appariement sur le score de propension, selon la méthode la mieux adaptée aux données. Ces analyses feront l'objet d'un Plan d'Analyse Statistique détaillé au préalable de leur réalisation,



mais rédigé une fois que les patients auront été inclus car la détermination des méthodes les mieux adaptées dépend de leur nombre et de leurs caractéristiques.

Les tests seront bilatéraux au seuil de 5%.

L'analyse reposant principalement sur des modèles à effets mixtes, il n'est pas prévu d'imputation des données manquantes, de par la difficulté accrue d'imputer convenablement des données longitudinales et du débat concernant le bénéfice d'une telle imputation par rapport à l'utilisation de modèles mixtes (Twisk J et al. *J Clin Epidemiol*, 2013, 66 :1022-1028).

Les 3 groupes (IRS antiandrogènes, sans traitement médicamenteux) seront décrits en utilisant la médiane, la moyenne, l'écart-type et la dispersion (écart interquartile), ou en termes de fréquence et de pourcentage (variables catégorielles);

Les estimations des paramètres d'intérêt pour l'analyse seront présentées avec leur intervalle de confiance à 95%. Une méthode exacte sera utilisée si nécessaire.

Les patients sous ISRS passant sous anti-androgène (switch) au cours de l'étude seront censurés à cette date. Si le switch intervient pendant la période de recrutement de l'étude, ils pourront être inclus dans le groupe de patients sous anti-androgène.

La principale mesure d'efficacité est le score quantitatif de l'intensité du désir sexuel au cours du temps. L'évolution de ce score sera analysée à l'aide d'un modèle linéaire mixte avec un effet sujet et une pente aléatoire. Un effet centre aléatoire pourra être ajouté au modèle s'il est trouvé significatif à l'aide d'un test de permutations. En outre, une analyse des trajectoires latentes sera effectuée pour identifier des classes de patients présentant des profils évolutifs similaires. Cette approche permettra de mieux comprendre les dynamiques sous-jacentes aux changements de l'intensité du désir sexuel et des symptômes associés.

Les covariables étudiées pour leur association avec les scores incluent: la durée antérieure du traitement, l'échec des traitements antérieurs (par exemple manque d'efficacité ou effets indésirables d'un traitement antérieur par antiandrogènes ayant nécessité un relais pour ISRS préalablement à l'inclusion), l'influence du type de paraphilie (pédophilie, exhibitionnisme, sadisme sexuel), les antécédents d'agressions sexuelles et non sexuelles antérieures, l'âge de début de la paraphilie, les caractéristiques socio-démographiques et cliniques (âge, niveau éducationnel, emploi et statut marital), et l'histoire personnelle et familiale d'autre trouble psychiatrique et de personnalité, des antécédents d'abus sexuels ou physiques, du fonctionnement cognitif, de l'utilisation de pornographie, de l'usage d'alcool ou de drogues illicites... Etant donné le nombre de variables étudiées, une pré-sélection sur des critères statistiques sera réalisée, et les modèles seront validés par des techniques de rééchantillonnage numérique (bootstrap).

Nous analyserons d'une part les scores quantitatifs de symptômes auto-évalués (intérêt sexuels et désir, pensées sexuelles ou fantasmes, activité sexuelle déviants et non déviants). Ces critères seront analysés de la même façon que le critère principal. D'autre part, les scores quantitatifs de l'intensité du désir sexuel et les symptômes auto-évalués seront dichotomisés, séparant les sujets sans intérêt sexuel, pensées ou activité paraphile (score égal à 0) qui définiront ceux bénéficiant d'un contrôle optimal de l'affection. Ces données seront analysées à l'aide de modèles linéaires généralisés à effets mixtes avec un lien logistique.

Le taux de rechute (la rechute étant définie comme l'occurrence d'une agression sexuelle quelconque parmi une série de conduites sexuelles prohibées par la loi comme le viol, les relations sexuelles avec un mineur, l'exhibitionnisme) et ses relations avec le type et la sévérité de la paraphilie et les autres caractéristiques seront analysées par modèle de régression à risque



proportionnel de Cox. L'incidence cumulée de rechute au cours du temps sera estimée et présentée, éventuellement de façon stratifiée ou ajustée sur des facteurs associés importants.

L'association des variations de l'impulsivité, de l'hypersexualité, des distorsions cognitives, de l'empathie, du déni, durant la période de suivi de 3 ans, sur les variations d'Intensité du désir et des symptômes sexuels sera analysée à l'aide de modèles mixtes de régression linéaire.

L'analyse des principaux indicateurs de sécurité mesurés par l'échelle CTCAE sera conduite selon les recommandations. La CTCAE distingue les événements en fonction de leur sévérité (grades 1-4 : léger, modéré, sévère et fatal respectivement). L'incidence des événements sera estimée et les facteurs de risque les plus fréquents seront examinés à l'aide de modèles de régression de Cox. Ces modèles seront utilisés pour tester le rôle de la durée du traitement, de l'observance, en contrôlant les variables socio-démographiques (âge, utilisation d'alcool ou de drogues illicites, pathologies somatiques comorbides ou traitements...), le type de paraphilie (pédophilie, exhibitionnisme, sadisme sexuel) et les traitements concomitants.

L'analyse des autres indicateurs (tension artérielle, fonction hépatique et rénale, profil lipidique, glycémie, numération sanguine, BMI, gynécomastie, ostéodensitométrie (Z scores), ECG (fréquence cardiaque, conduction cardiaque) sera conduite avec la même stratégie.

Les autres mesures, dépression, tentatives de suicide, activité sexuelle non déviante seront décrites ainsi que leur évolution durant la période de suivi de 3 ans.

## Analyses exploratoires

Des analyses exploratoires seront conduites dans un second temps pour évaluer la variation du critère principal chez les patients observants et non-observants, et l'effet des traitements associés (thérapie cognitivo-comportementale ou psychothérapie). Ces analyses utiliseront des modèles causaux (modèles structuraux marginaux, modèles structuraux emboîtés [G-estimation] ou modèles de stratification principale). Le modèle sera déterminé en fonction des données disponibles, et de la vérification (ou non) des hypothèses sous-jacentes aux différents modèles.

Une étude descriptive de la population comprendra : à l'inclusion

- date et lieu de naissance,
- taille et poids (l'IMC sera calculé),
- le plus haut niveau d'éducation atteint,
- le type d'emploi actuel et passé,
- le fait de vivre seul ou avec un partenaire, le nombre d'enfants (âge et sexe),
- les antécédents personnels et familiaux (1<sup>er</sup> et 2<sup>nd</sup> degré) de troubles psychiatriques et de troubles paraphiles ou d'antécédents judiciaires,
- le type et les caractéristiques cliniques des paraphilies,
- l'âge d'apparition des paraphilies et des premiers fantasmes déviants ou paraphiles,
- le nombre et le type d'infractions sexuelles ou non sexuelles précédentes ayant été condamnées,
- les traitements antérieurs reçus pour les troubles paraphiles (type de médicament, dose par jour, date de la première utilisation et d'interruption le cas échéant, la raison du changement de dose ou de traitement le cas échéant),
- traitement actuel reçu (type de médicament, dose par jour, date de la première utilisation)
- maladies et traitements somatiques concomitants (en particulier épilepsie, démence, retard mental, traumatisme cérébral avec perte de connaissance avec âge de survenue, maladie neurologique, méningiome, syndrome métabolique),



- utilisation de la pornographie (oui / non, le type (déviant ou non) ; âge de 1<sup>ère</sup> exposition, la fréquence d'utilisation par mois et l'âge de la première utilisation),
- les antécédents de comportement sexuel non déviant (le cas échéant), l'âge du premier rapport sexuel, l'âge de la puberté, l'existence d'une intervention chirurgicale pour phimosis ou ectopie testiculaire et l'âge de survenue de celle ci
- la consommation d'alcool et la consommation de drogue illicite (âge de début, quantité par jour, type)

## 10.2 HYPOTHESE DE CALCUL DU NOMBRE DE SUJETS NECESSAIRES ET RESULTAT

Un échantillon de 75 patients est prévu dans le groupe ISRS. Cette taille d'échantillon permet de construire des modèles de régression avec 10 à 15 variables que l'on considère habituellement comme suffisamment robustes (règle de 10 patients par variable pour les modèles de régression linaire, par exemple).

Un échantillon de 25 sujets (correspondant à 75 personnes-années) dans le groupe traité par antiandrogènes, permettra d'obtenir une estimation suffisamment précise de l'incidence des effets indésirables. Plus précisément, la largeur de l'intervalle de confiance à 95% sera de 12% (±6%) pour une incidence annuelle de 20%.

Un échantillon de 100 patients sera inclus dans le groupe ne recevant pas de traitement pharmacologique.

## Proposition:

La taille de l'échantillon proposée pour l'étude est basée sur des considérations pratiques et empiriques, en l'absence de littérature spécifique pouvant guider une estimation précise. Compte tenu de la nature observationnelle de l'étude, de la population limitée, des réticences probables à participer à l'étude, ainsi que du manque de littérature solide dans le domaine, un échantillon de 75 patients est prévu dans le groupe traité par ISRS. Cet échantillon permettra d'explorer les relations entre les variables d'intérêt dans le contexte de notre étude.

Un échantillon de 25 sujets dans le groupe traité par antiandrogènes, correspondant à 75 personnes-années, permettra d'obtenir une estimation raisonnablement précise de l'incidence des effets indésirables. Plus précisément, la largeur de l'intervalle de confiance à 95 % sera de  $\pm 6$  % pour une incidence annuelle de 20 %.

Enfin, un échantillon de 100 patients sera inclus dans le groupe ne recevant pas de traitement pharmacologique, avec pour objectif de garantir une représentation adéquate de cette population et de permettre des comparaisons significatives avec les groupes traités.

Bien que la taille de l'échantillon proposée soit basée sur des considérations pratiques et empiriques, nous estimons qu'elle est appropriée pour atteindre les objectifs de l'étude, compte tenu des contraintes déjà mentionnées. Cependant, il est important de noter que les résultats devront être interprétés avec prudence, en raison de l'absence de données antérieures permettant de fournir une estimation plus précise de la puissance statistique.

## 11. CONTRÔLE ET ASSURANCE DE LA QULITÉ



## 11.1 ORGANISATION GÉNÉRALE

Le promoteur doit s'assurer de la sécurité et du respect des personnes qui ont accepté de participer à la recherche. Il doit mettre en place un système d'assurance qualité permettant de surveiller au mieux le déroulement de la recherche dans les centres investigateurs.

A cet effet le promoteur définira une stratégie d'ouverture des centres et pourra le cas échéant mettre un place un contrôle qualité des données.

### 11.2 Stratégie d'ouverture des centres

La stratégie d'ouverture des centres sera déterminée avant le démarrage de la recherche.

#### 11.3 Contrôle qualité des données

Un Attaché de Recherche Clinique (ARC) mandaté par le promoteur s'assurera de la bonne réalisation de la recherche, du recueil des données générées par écrit (pour l'ECG par exemple) ou électroniquement, de leur documentation, enregistrement et rapport, en accord avec les Procédures Opératoires Standard mises en application au sein de la DRCI.

L'investigateur et les membres de son équipe acceptent de se rendre disponibles lors des visites de Contrôle de qualité effectuées à intervalles réguliers par l'Attaché de Recherche Clinique.

#### 11.4 Cahier d'observation

## <u>CRF électronique</u>:

Toutes les informations requises par le protocole doivent être consignées dans les cahiers d'observation électronique. Les données devront être recueillies au fur et à mesure qu'elles sont obtenues, et enregistrées dans ces cahiers de façon explicite. Chaque donnée manquante devra être codée.

Ce cahier d'observation électronique sera mis en place dans chacun des centres grâce à un support Internet de recueil des données. Un document d'aide pour l'utilisation de cet outil sera fourni aux investigateurs.

Le remplissage du cahier d'observation via internet par l'investigateur permet ainsi à l'ARC de visualiser rapidement et à distance les données. L'investigateur est responsable de l'exactitude, de la qualité et de la pertinence de toutes les données saisies. De plus, lors de leurs saisies, ces données sont immédiatement vérifiées grâce à des contrôles de cohérence. L'investigateur doit valider toute modification de valeur dans le CRF. Une justification peut éventuellement être intégrée en commentaire.

Une impression papier sera demandée en fin d'étude, authentifiée (datée et signée) par l'investigateur. L'original de ce document sera archivé par le promoteur. Une copie du document authentifié devra être archivée par l'investigateur.

#### 11.5 Gestion des non conformités

Tout évènement survenant suite au non-respect du protocole, des procédures opératoires standardisées, ou des dispositions législatives et réglementaires en vigueur par un investigateur ou toute autre personne impliquée dans la conduite de la recherche doit faire l'objet d'une déclaration de non-conformité au promoteur.



Ces non conformités seront gérées conformément aux procédures du promoteur.

#### 11.6 Audit

Les investigateurs s'engagent à accepter les audits d'assurance qualité effectués par le promoteur ainsi que les inspections effectuées par les autorités compétentes. Toutes les données, tous les documents et rapports peuvent faire l'objet d'audits et réglementaires sans que puisse être opposé le secret médical.

Un audit peut être réalisé à tout moment par des personnes mandatées par le <u>promoteur</u> et indépendantes des responsables de la recherche. Il a pour objectif de s'assurer de la qualité de la recherche, de la validité de ses résultats et du respect de la loi et des règlementations en vigueur.

Les personnes qui dirigent et surveillent la recherche acceptent de se conformer aux exigences du promoteur en ce qui concerne un audit.

L'audit pourra s'appliquer à tous les stades de la recherche, du développement du protocole à la publication des résultats et au classement des données utilisées ou produites dans le cadre de la recherche.

## 11.1.6 Engagement de responsabilités de l'Investigateur Principal

Avant de démarrer la recherche, chaque investigateur fournira au représentant du promoteur de la recherche son curriculum vitæ personnel actualisé, daté de moins d'un an et signé, comportant son numéro RPPS. Le CV devra comprendre les participations antérieures à des recherches et les formations liées à la recherche clinique.

Chaque investigateur s'engagera à respecter les obligations législatives et réglementaires et à mener la recherche conformément à la réglementation, en respectant les termes de la déclaration d'Helsinki en vigueur.

L'investigateur principal de chaque centre participant signera un engagement de responsabilités (document type DRCI) qui sera remis au représentant du promoteur.

Les investigateurs et leurs collaborateurs signeront un formulaire de délégation de fonctions précisant le rôle de chacun et fourniront leur CV.

## 12. ASPECTS ETHIQUES ET LEGAUX

## 12.1 MODALITÉS D'INFORMATION ET DE RECUEIL DU CONSENTEMENT DES PERSONNES SE PRÊTANT A LA RECHERCHE

Le patient (si nécessaire son curateur) sera informé par son psychiatre traitant ou le médecin investigateur des risques et bénéfices de l'étude et signera un consentement écrit et éclairé s'il souhaite participer après avoir lu la note d'information et avant l'inclusion. Il recevra un double du consentement et une copie du formulaire d'information.

Conformément à l'article L1122-1-1 du Code de la santé publique, aucune recherche à risque et contraintes minimes impliquant la personne humaine ne peut être pratiquée sur une personne sans son consentement libre et éclairé, et exprès après que lui a été délivrée l'information prévue à l'article L. 1122-1 du même code.



Un délai de réflexion de 7 jours si vous voulez est laissé à la personne entre le moment où elle est informée et celui où elle signe le formulaire de consentement.

Le consentement libre, éclairé et écrit de la personne est recueilli par l'investigateur principal, ou par un médecin qui le représente ou par la personne qualifiée avant l'inclusion de la personne dans la recherche lors de l'inclusion.

La note d'information et une copie du formulaire de consentement daté et signé par la personne qui se prête à la recherche ainsi que par l'investigateur ou le médecin qui le représente ou la personne qualifiée, sont remis à la personne préalablement à sa participation à la recherche.

En outre, l'investigateur précisera dans le dossier médical de la personne la participation de celleci à la recherche, les modalités de recueil de son consentement [ou du consentement de toute autre personne dans les cas prévus aux articles L. 1122-1-1 à L. 1122-2 du CSP] ainsi que les modalités de la délivrance de l'information en vue de le recueillir. Il conserve un exemplaire original du formulaire du recueil du consentement de la personne daté et signé.

# 12.2 INTERDICTION POUR LA PERSONNE DE PARTICIPER A UNE RECHERCHE OU PERIODE D'EXCLUSION PRÉVUE A L'ISSUE DE LA RECHERCHE, LE CAS ÉCHÉANT

Pendant sa période de participation à la recherche le patient ne peut pas participer à un autre protocole de recherche impliquant la personne humaine sans en avoir parlé avec le médecin qui le suit dans le cadre de la recherche.

A la fin de la participation du patient, aucune période d'exclusion n'est définie dans le cadre de cette recherche.

Pendant la durée de sa à la recherche le patient peut participer simultanément à un autre protocole de recherche impliquant la personne humaine

#### 12.3 INDEMNISATION DES SUJETS

Non applicable car soins courants

Remboursement des frais exposés

Aucune indemnisation n'est prévue dans le cadre de cette étude

#### 12.4 OBLIGATIONS LÉGALES

#### 12.4.1 Rôle du promoteur

Le Groupe Hospitalier Universitaire Paris – Psychiatrie & Neurosciences (GHU Paris) est le promoteur de cette recherche et par délégation la Délégation à la Recherche Clinique et à l'Innovation (DRCI) en assure les missions, conformément à l'article L.1121-1 du code de la santé publique. Le GHU PARIS se réserve le droit d'interrompre la recherche à tout moment pour des raisons médicales ou administratives dans cette éventualité, une notification sera fournie à l'investigateur.



## 12.4.2 Demande d'avis au Comité de Protection des Personnes (CPP)

Le GHU Paris en tant que promoteur obtient pour la recherche à risque et contraintes minimes, préalablement à sa mise en œuvre l'avis favorable du CPP concerné, dans le cadre de ses compétences et conformément aux dispositions législatives et réglementaires en vigueur.

# 12.4.3 Information de l'Agence Nationale de Sécurité du Médicament et des produits de santé (ANSM)

Le promoteur transmettra à l'ANSM le résumé de la recherche ainsi que l'avis favorable du Comité de Protection des Personnes.

### 12.4.4 Modifications de la recherche

Toute modification substantielle apportée au protocole par l'investigateur coordonnateur, devra être transmise au promoteur pour approbation. Après cet accord, le promoteur devra obtenir préalablement à sa mise en œuvre un avis favorable du CPP.

La note d'information et le formulaire de consentement pourront être révisés si nécessaire, notamment en cas de modification substantielle de la recherche ou de la survenue d'effets indésirables.

### 13. FINANCEMENT ET ASSURANCE

#### **13.1 SOURCE DE FINANCEMENT**

PHRC national

### 13.2 ASSURANCE

Le Promoteur, souscrit pour toute la durée de la recherche une assurance garantissant sa propre responsabilité civile ainsi que celle de tout médecin impliqué dans la réalisation de la recherche. Il assure également l'indemnisation intégrale des conséquences dommageables à la recherche pour la personne qui s'y prête et ses ayants droit, sauf preuve à sa charge que le dommage n'est pas imputable à sa faute ou à celle de tout intervenant, sans que puisse être opposé le fait d'un tiers ou le retrait volontaire de la personne qui avait initialement consenti à se prêter à la recherche.

Le Groupe Hospitalier Universitaire Paris – Psychiatrie & Neurosciences (GHU Paris) a pris une assurance auprès de la compagnie Relyens Mutual Insurance (Police N°163543) garantissant sa responsabilité civile ainsi que celle de tout intervenant (médecin ou personnel impliqué dans la réalisation de la recherche), conformément à l'article L.1121-10 du CSP.

## 14. RÉGLES RELATIVES A LA PUBLICATION

Le GHU Paris devra obligatoirement être mentionné dans les affiliations du ou des auteurs des publications qui résulteront de cette recherche et mentionner le promoteur (GHU Paris /DRCI) et la source de financement si votre projet résulte d'un appel d'offres (par exemple le PHRC national ou régional), et nous en adresser un exemplaire (cf. ci-dessous les modalités d'affiliation et de mention du promoteur et du financeur).



## 14.1 MENTION DE L4AFFILIATION DU GHU PARIS POUR LES PROJETS PROMUS OU GÉRÉS PAR LE GROUPE HOSPITALIER UNIVERSITAIRE PARIS – PSYCHIATRIE & NEUROSCIENCES

- Si un auteur a plusieurs affiliations, l'ordre dans lequel sont citées les institutions (GHU Paris, Université, INSERM...) n'a pas d'importance
- Chacune de ces affiliations doit être identifiée par une adresse séparée par un point-virgule (;).

# 14.2 MENTION DU PROMOTEUR GHU PARIS (DRCI) DANS LES « ACKNOWLEDGMENTS » DU MANUSCRIT

" The sponsor was GHU Paris/DRCI"

# 14.3 MENTION DU FINANCEUR DANS LES « ACKNOWLEDGMENTS » DU MANUSCRIT

"The study was funded by a grant from Programme Hospitalier de Recherche Clinique - PHRC 2015 (Ministère de la Santé)"

## 15. BIBLIOGRAPHIE

• Echelle PATHOS/ (PATHOS Scale, Carnes et al., 2012; traduction française : L Karila, Thibaut, Acuna-Vargas et al.) **Autoévaluation** 

L'échelle PATHOS (<u>P</u>reoccupied, <u>A</u>shamed, <u>T</u>reatment, <u>H</u>urt others, <u>O</u>ut of control, <u>S</u>ad) comprend 6 items (réponses par oui ou non). Durée : 1 min. Cet instrument sera utilisé pour classer les patients en hypersexuels ou non. L'échelle PEACCE a inclus 92,6% de l'aire sous la courbe, et a permis de distinguer des hommes présentant une hypersexualité, en utilisant un cut off de 3, avec une sensibilité de 88.3% et une spécificité de 81.6% (échelle diagnostique).

• Le questionnaire de personnalité PDQ-4+ (Hyler, 1994) traduction française Bouvard., 2011) **Autoévaluation** 

Le questionnaire de personnalité permet une autoévaluation des troubles de personnalité à l'aide de 99 questions Administration : 10-15 minutes.

• Echelle d'intensité du désir et des symptômes sexuels (<u>échelle d'auto-évaluation</u> utilisée pour la mesure des comportements sexuels déviants et non déviants). **Autoévaluation** 

Cette échelle mesure 3 aspects du comportement sexuel (Rösler and Witztum, NEJM, 1998, modifié de Bancroft et al., 1974)

Le comportement sexuel inclut à la fois un comportement fantasmé et déclaré. L'excitation sexuelle auto-rapportée (réponse subjective) concerne la manière avec laquelle un individu appréhende et rapporte son état émotionnel en ce qui concerne l'excitation sexuelle. La plupart des chercheurs demandent aux participants de coter leur excitation sexuelle en utilisant des items de type Likert. L'excitation sexuelle subjective et la perception de la réponse génitale sont fortement et positivement corrélées chez les femmes (Slob, Bax, Hop, Rowland, & van der Werff ten Bosch, 1996) comme chez les hommes (Rowland & Heiman, 1991; pour des méta analyses récentes, voir Chivers et al., 2010).

L'échelle d'intensité du désir et des symptômes sexuels (ISDSS) va permettre de mesurer 3 types d'intérêt et comportements sexuels :



(1) intérêt sexuel et désir, les sujets devront indiquer la nature, l'intensité et la fréquence de leurs pensées et désirs sexuels, durant le mois précédent la visite (d'aucune pensée sexuelle jusqu'à pensées très fréquentes avec pulsions sexuelles intenses); (2) pensées sexuelles ou fantasmes, les sujets devront décrire leurs fantasmes érotiques les plus intenses et prolongés, et décrire l'objet de ce fantasme (enfant ou adulte, homme, femme ou les 2, etc.), son intensité (d'aucune excitation à excitation maximale) et la fréquence du fantasme par semaine, durant le mois précédant la visite, et finalement (3) mesure de l'activité sexuelle, les sujets devront renseigner le nombre de fois par semaine où il se seront masturbés, le nombre de fois où ils auront entrepris (et déclaré) un acte conduisant à un orgasme, et la nature et le nombre d'incidents de comportement anormal (s'il y en a) dans le mois précédent. Chacun des trois types de comportement sera coté selon une échelle de type Likert allant de 0 à 8, et la moyenne des trois scores sera utilisée. Un score de 1 indique une excitation sexuelle nulle ou minime, et une absence de fantasme ou comportement sexuel, alors qu'un score de 8 correspond à une excitation et un comportement sexuels incontrôlés. Les études test-retest de cette autoévaluation ont montré une fiabilité satisfaisante pour des pensées sexuelles dans des limites acceptables (Tennent et al., 1974). Pour Tennent et al. (1974), pour ce qui concerne le comportement sexuel déclaré, l'approche la plus simple est le décompte de la fréquence des comportements spécifiques.

Les activités sexuelles conventionnelles ou non seront cotées séparément. De plus, les scores de comportement sexuel déviant seront séparés entre les sujets sans (score égal à 0) intérêt sexuel déviant, pensées ou activités et les autres. Ceux présentant un score de 0 seront considérés comme bénéficiant d'un contrôle thérapeutique optimal de leur affection.

La durée totale du test ne devrait pas dépasser 10 minutes.

- Evaluation du risque de violence sexuelle et non sexuelle
- Echelle actuarielle de type statique d'évaluation du risque de récidive à l'inclusion :

Static 99 (Hanson et Thornton, 1999; traduction française: Ducro et Pham, 2006) Il s'agit d'un outil d'évaluation de type actuariel, qui permet l'évaluation du score de récidive selon 4 niveaux, de faible à élevé, conduisant à une estimation de probabilité de récidive à 5 ans de 6 %, 11 %, 30 % et 39 %. La passation de la Static-99 repose sur le casier judiciaire du sujet ainsi que toutes sources d'information possible. Cet outil présente de bonnes qualités prédictives pour la récidive sexuelle (AUC 0,72) mais également pour la récidive violente y compris sexuelle. Sa validité prédictive varie en fonction du type de délit, modérée pour l'inceste (0,74), le viol (0,71), marginale pour les pédophiles extra-familiaux (0,65), mais très bonne pour la récidive violente chez les auteurs d'inceste (0,92), modérée auprès de pédophiles extra-familiaux (0,87); elle est adaptée aux adultes de sexe masculin de plus de 18 ans, est évaluée sur dossier pour un temps de passation d'environ 10 minutes.



## ANNEXE I

## Règles de codage de la Statique-99

| Facteur de risque | Codes | | Score |
|---|---|---|---|
| Infractions sexuelles antérieures | Accusations | Condamnations | |
| (Mêmes règles que pour l'ERRRS) | | | |
| | Aucune | Aucune | 0 |
| | 1-2 | 1 | 1 |
| | 3-5 | 2-3 | 2 |
| | 6 + | 4 + | 3 |
| Prononcés de peine antérieurs | 3 ou moins | | 0 |
| (non comprise l'infraction répertoriée) | 4 ou plus | | 1 |
| Condamnations pour infractions | Non | | 0 |
| sexuelles sans contact | Oui | | 1 |
| Infractions de violence non sexuelle | Non | | 0 |
| répertoriées | Oui | | 1 |
| Infractions de violence non sexuelle | Non | | 0 |
| antérieures | Oui | | 1 |
| Au moins une victime sans lien de | Non | | 0 |
| parenté avec le délinquant | Oui | | 1 |
| Au moins une victime qui était un | Non | | 0 |
| inconnu | Oui | | 1 |
| Au moins une victime du sexe | Non | | 0 |
| masculin | Oui | | 1 |
| Jeune | 25 ans ou plus | | 0 |
| | 18 - 24,99 ans | | 1 |
| Célibataire | Le délinquant a-t- | | |
| | pendant au moins | deux ans avec son | |
| | amant? (homme o | ou femme) | |
| | Oui | | 0 |
| | Non | | 1 |
| Score total | Faire la somme d | es scores obtenus | |
| | pour différents fa | cteurs de risque | |

## TRANSFORMATION DES SCORES OBTENUS SUR LA STATIQUE-99 EN CATÉGORIES DE RISQUE

| Score | Catégorie de risque |
|-----------|---------------------|
| 0,1 | Faible |
| 2,3 | Faible-moyen |
| 4,5 | Moyen-élevé |
| 6 ou plus | Élevé |

6 plus High



## Tableau 3 — Items de la Statique-99

- Infractions sexuelles antérieures (accusations ou condamnations);
- Prononcés de peine(s) antérieurs;
- Condamnations pour infractions sexuelles sans contact;
- Infractions de violence non sexuelle répertoriées;
- Infractions de violence non sexuelle antérieures;
- Au moins une victime sans lien de parenté avec le délinquant;
- Au moins une victime qui était un inconnu;
- Au moins une victime de sexe masculin :
- Jeune :
- Célibataire.

## Facteur 1 : Prédicteurs stables

Influences sociales importantes

Amants / Partenaires intimes;

Identification émotive aux enfants;

Hostilité envers les femmes;

Solitude / Isolement / Rejet social en général;

Manque d'intérêt à l'égard des autres.

Problèmes sur le plan de l'intimité

Amants / partenaires intimes;

Identification émotive aux enfants;

Hostilité envers les femmes ;

Solitude / Isolement / Rejet social en général;

Manque d'intérêt à l'égard des autres.

Maîtrise de soi sur le plan sexuel

Libido / Préoccupations sexuelles;

Recours au sexe comme mécanisme d'adaptation;

Intérêts sexuels déviants.

Attitudes tolérantes à l'égard de l'agression sexuelle

Droit au sexe:

Attitudes favorables face au viol;

Attitudes propices à l'agression d'enfants.

- Coopération dans le cadre de la surveillance
- Maîtrise de soi en général

Gestes impulsifs;

Faibles aptitudes cognitives pour la résolution de problèmes ;

Émotions négatives / Hostilité.

### Facteur 2 : Prédicteurs aigus

- Accès aux victimes;
- Effondrement émotionnel :
- Écroulement des soutiens sociaux ;
- Hostilité;
- Consommation d'alcool ou de drogue;
- Préoccupations sexuelles ;
- Refus de surveillance;
- Facteur unique.
  - STABLE-2007 (Eher, Matthes, Schilling, Haubner-MacLean et Rettenberg, 2011) traduit et validé en français par T Pham Université de Mons Belgique



Il s'agit d'une évaluation des risques de récidive sexuelle.

Les facteurs de risque dits dynamiques sont des caractéristiques durables (mais potentiellement modifiables) d'un délinquant, généralement formulées en termes de traits ou d'états psychologiques, qui sont associées à la récidive.

Ces caractéristiques associées à la récidive sexuelle sont par exemple : Les intérêts sexuels déviants, les fréquentations criminelles et l'instabilité conjugale. Bien qu'ils soient modifiables, les facteurs dynamiques stables sont, conformément à leur appellation, assez stables.

Durée de passation : entre 60 et 120 minutes, voire plus. Hétéroévaluation via entretien semidirectif.

La formation à ces échelles a déjà été assurée par le Dr Ducro pour l'ensemble des centres investigateurs.

• Inventaire de Dépression de Beck, Beck Depression Inventory (BDI-II) (<u>Beck et al. 1996</u>; Traduction française, Bourque et al.,1982) **Autoévaluation** 

La version proposée est une version à 13 items dérivant de la version à 21 items, validée en français. Il s'agit d'un <u>auto-questionnaire</u>. Chaque item exprime 4 propositions, qui reflètent l'intensité de symptômes dépressifs allant du neutre (Je ne me sens pas triste) à sévère (je suis si triste ou malheureux que je ne peux plus le supporter). Chaque proposition se voit attribuer un score entre 0 et 3, et la somme de ces valeurs (entre 0 et 39) fournit un score global qui permet d'effectuer la comparaison du sujet avec lui-même au cours du temps ou avec d'autres. Les items explorent des mesures de symptômes dépressifs, cognitifs, affectifs, somatiques, et végétatifs. L'avantage de cet outil est sa bonne consistance interne, avec un coefficient alpha de Cronbach variant entre 0.89 et 0.93, son excellente validité de contenu, sa sensibilité au changement, et finalement sa capacité à discriminer entre les sujets déprimés et non déprimés (Beck et al., 1998; <u>Dozois et al. 1998</u>). La durée totale de ce test n'excède pas 10 minutes.

• Echelle d'intentionnalité suicidaire de Beck, Beck Scale for Suicide Ideation (BSSI) (Beck et al., 1979) **Autoévaluation** 

Il s'agit d'un outil <u>d'auto-évaluation</u> validé en français. Il consiste en 21 items, et peut être utilisé pour détecter et mesurer la sévérité des idées et comportements suicidaires (19 premiers items), les 2 dernières questions évaluant le nombre de tentatives de suicide antérieures et l'intention de mourir associée à la dernière tentative, les 2 derniers items ne sont pas comptés dans le score. Chacun des 19 premiers items est scoré de 0 à 2 (score maximum 38). Le psychiatre détermine ainsi, si possible, le risque suicidaire durant une visite, la conduite à tenir (hospitalisation, initiation d'un traitement spécifique, et ces éléments sont enregistrés et inclus dans l'analyse finale). En utilisant un cut off de 24, le BSSI présente d'excellentes sensibilité (100%) et spécificité (90%) pour prédire l'hospitalisation parmi des patients suicidaires avec une valeur prédictive positive globale de 71% (Cochrane-Bink et al., 2000). Durée totale du test environ 10 minutes.

#### Hypersexualité

L'Inventaire du comportement sexuel compulsif ou Compulsive Sexual Behavior Inventory (CSBI) sera utilisé pour évaluer la sévérité de l'hypersexualité (CSBI-22; Miner et al., 2007; Traduction et validation française réalisée par notre équipe). Le CSBI permettra de mesurer les changements. Chacun des 22 items est coté sur une échelle en 5 points, allant de jamais à très fréquent, avec une fiabilité de 0.86; l'échelle contrôle est représentée par les items 1 à 13, et l'échelle violence de 14 à 22. Les scores les plus bas indiquent une addiction sexuelle plus faible. La durée du test est d'environ 10 minutes. **Autoévaluation** 



• Echelle de qualité de vie (SF-36): SF-36 (Medical Outcome Study 36 – Item Short Form Health Survey) (Ware and Sherbourne, 1992; Traduction française, Leplege et al., 1995) Ce questionnaire de 36 items évalue 8 dimensions (chacune étant cotée de 0 à 100, un score plus élevé indiquant une meilleure santé) afin de mesurer la qualité de vie en lien à la santé physique et psychique du point de vue du patient. La durée du test est d'environ 10 minutes. **Autoévaluation** 

• Evaluation des effets indésirables : utilisation de la version 4.0 des Critères de Terminologie Communs des événements indésirables, Common Terminology Criteria for Adverse Events (CTCAE) (<a href="http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE">http://evs.nci.nih.gov/ftp1/CTCAE/CTCAE</a> 4.03 2010-06-14 OuickReference 5x7.pdf). (Pour revue, voir Edwards and Aronson, 2000)

Les critères CTCAE permettent de distinguer les événements en fonction de leur sévérité (grades 1-4 : léger, modéré, sévère, et fatal, respectivement). **Autoévaluation** 

- Echelle d'évaluation brève de l'observance : Brief Adherence Rating Scale (BARS scale) (Byerly et al., 2008) sauf chez ceux ne recevant pas de traitement L'échelle BARS a été récemment développée, il s'agit d'un outil administré par le clinicien destiné à évaluer l'observance, à l'aide de 3 questions concernant la connaissance qu'a le patient de son traitement et les épisodes d'oublis de prises, selon le schéma suivant :
  - 1. Nombre de doses de traitement prescrites par jour
- 2. Nombre de jours au cours du mois précédent au cours desquels le patient n'a pas pris la dose prescrite
- 3. Nombre de jours au cours du mois précédent au cours desquels le patient a pris une dose moindre que celle prescrite

Une échelle visuelle analogique est utilisée pour évaluer la proportion de doses prises durant le mois précédent (0–100%). La cotation par échelle visuelle analogique est la mesure clé du la cotation par la BARS. Elle a pu montrer une bonne sensibilité et une bonne spécificité. En ce qui concerne l'adhérence en elle-même, la BARS semble être le meilleur choix, et a été étudiée de manière extensive dans la schizophrénie, pathologie au cours de laquelle l'observance est un problème majeur (Acosta et al., 2012). La durée du test est d'environ 1 minute **Autoévaluation** 

• Échelle d'impulsivité de Barratt (BIS-11 ; Patton et al., 1995. Traduction et validation française : F.J. Baylé, H. Caci, E.S. Barratt, J.D. Guelfi, R. Jouvent, J.P. Olié

L'échelle est un questionnaire en auto-évaluation conçu pour évaluer le concept personnalité / comportement de l'impulsivité.

La version actuelle de l'échelle Barratt Impulsiveness Scale (BIS-11; Patton et al., 1995) est composée de 30 éléments/items (décrivant les comportements et préférences communs impulsifs ou non impulsifs (pour les éléments à scores inversés)) sur une échelle de Likert (1 à 4) qui permettent d'évaluer de multiples facettes de l'impulsivité, dont l'attention, l'impulsivité motrice, l'autocontrôle (planification et réflexion), la complexité cognitive (appréciation des tâches réflexives), la persévérance (stabilité du mode de vie) et l'instabilité

cognitive (fuite des idées). Le questionnaire BIS version 11. Le BIS-11 reste la mesure d'impulsivité la plus utilisée aujourd'hui et le modèle sur lequel elle est basée (trois composantes principales de l'impulsivité : motrice, attentionnelle et non planifiée). Durée totale 5 à 10 minutes. Autoévaluation.



# 15.1 ECHELLES D'AGRESSION ET DE VIOL, MOLEST AND RAPE SCALES (Bumby KM, 1996) (Traduction française : T Pham)

Les échelles MOLEST et RAPE sont destinées à évaluer les distorsions cognitives respectivement des agresseurs et auteurs de viols d'enfants. Les résultats indiquent que ces mesures sont prometteuses tant en clinique que pour la recherche, présentant une validité et une consistence interne fortes, une bonne validité convergente et discriminative, sans biais de désirabilité sociale, et sont utiles pour évaluer l'efficacité sur le plan de la restructuration cognitive d'un traitement. De plus, les distorsions cognitives des agresseurs sexuels évaluées à l'aide de ces échelles ont montré un lien avec le nombre de victimes et la durée du comportement d'agression sexuelle. La durée du test est d'environ 15 minutes. **Autoévaluation** 

# 15.2 L'ECHELLE D'EMPATHIE (BES Basic Empathy Scale) (Joliffe et Farrington., 2006 ; Traduction française D'Ambrosio et al. 2008)

L'amélioration des capacités d'empathie est un objectif commun des traitements des agresseurs sexuels qui pourrait influencer le maintien du comportement sexuel déviant, et qui est difficile à évaluer. La BES a été validée pour l'évaluation de l'empathie dans plusieurs études conduites auprès de violeurs et agresseurs d'enfants. Elle inclut 20 items dont on addditionne les scores qui vont de 1 à 5. La durée du test est d'environ 10 minutes. **Autoévaluation** 

# 15.3 GRILLE D'EVALUATION DU DENI ET DE LA MINIMISATION (McKibben A, Aubut J, Dassylva B (1995). Grille d'évaluation du déni et de la minimisation.

Cet outil évalue le déni en relation avec les faits, la responsabilité, les conséquences pour la victime, les problèmes personnels liés aux faits, les fantasmes sexuels déviants, la nécessité d'un traitement lié à un comportement sexuel. (Les réponses vont de 1: déni total 5: entièrement d'accord). Les 6 scores seront additionnés puis le total divisé par 6 pour obtenir un score moyen de déni. La durée du test est d'environ 10 min. **Autoévaluation** 

# 15.4 QUESTIONNAIRE D'HISTOIRE TRAUMATIQUE, Trauma History Questionnaire (THQ) (Hooper et al., 2011 traduction française : Jehel et al., 2000)

Le THQ est une <u>auto-évaluation</u> en 24 points qui examine les expériences d'événements potentiellement traumatiques tels que la criminalité, une catastrophe naturelle, et l'agression sexuelle et physique à l'aide d'un format oui/non. Pour chaque événement approuvé, les sujets sont invités à préciser la fréquence de l'événement ainsi que leur âge au moment de sa survenue. Le THQ peut être utilisé dans les milieux cliniques et de recherche. Il dispose d'une bonne fiabilité test-retest sur une période de plusieurs semaines (r = 0,60 à 1,00 pour les événements individuels, vécus personnellement). Dans la présente étude, les réponses à la THQ seront utilisées pour évaluer l'étendue des agressions et des abus que les sujets ont rapportés dans leurs sphères physiques et sexuelles, ainsi que des antécédents de maladie potentiellement mortelle avant de développer des troubles paraphiliques. Les réponses sous forme d'auto-évaluation seront suivies d'un entretien en face-à-face pour recueillir des détails supplémentaires. L'existence d'un traumatisme sexuel sera évaluée par trois questions (par exemple, "Quelqu'un vous a-t-il jamais forcé à avoir des rapports sexuels, oraux ou anaux contre votre volonté ?"). Ces items seront additionnés, avec des scores pouvant aller de 0 à 3. L'existence d'un traumatisme physique sera évaluée par quatre questions (par exemple, "Quiconque incluant un membre de votre famille vous a-t-il déjà attaqué sans arme et sérieusement blessé". Ces items seront également additionnés,



fournissant des scores de 0 à 4. La durée du test est d'environ 10 min. Autoévaluation

# 15.5 LE QUESTIONNAIRE AUDIT C POUR PREPARER LES CONSOMMATIONS EXCESSIVES D'ALCOOL DANS TOUTES LES ETUDES PUBLIEES

## Le questionnaire AUDIT-C

Un score  $\geq$  3 chez la femme et  $\geq$  4 chez l'homme doit faire évoquer un mésusage.

Un score ≥ 10 dans les deux sexes doit faire évoquer une dépendance. La durée de passation est de 1 min. **Autoévaluation** 

- 1. À quelle fréquence vous arrive-t-il de consommer des boissons contenant de l'alcool ?
- (0) Jamais
- (1) 1 fois par moi ou moins
- (2) 2 à 4 fois par mois
- (3) 2 à 3 fois par semaine
- (4) Au moins 4 fois par semaine
- 2. Combien de verres standard buvez-vous au cours d'une journée ordinaire où vous buvez de l'alcool ?
- (0) 1 ou 2
- (1) 3 ou 4
- (2) 5 ou 6
- (3) 7 à 9
- (4) 10 ou plus
- 3. Au cours d'une même occasion, à quelle fréquence vous arrive-t-il de boire six verres standard ou plus ?
- (0) Jamais
- (1) Moins d'une fois par mois
- (2) Une fois par mois
- (3) Une fois par semaine
- (4) Tous les jours ou presque

## **15.6 MOCA**

Evaluation rapide par hétéroquestionnaire des fonctions cognitives

Le MoCA (Nasreddine et al., 2005) a pour objectif essentiel le dépistage des personnes qui vivent une atteinte neurocognitive de légère à sévère.

Nasreddine, Z. S., Phillips, N. A., Bédirian, V., Charbonneau, S., Whitehead, V., Collin, I., ...et Chertkow, H. (2005). The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. *Journal of the American Geriatrics Society*, 53(4), 695-699.

Le MoCA est un outil de dépistage de l'atteinte neurocognitive et il est dédié principalement au dépistage de l'atteinte plus légère. Le MoCA est un questionnaire à réponses courtes incluant quelques tâches que doit accomplir la personne. Les éléments évalués sont regroupés en six sous-sections : mémoire à court terme, habiletés visuospatiales, fonctions exécutives, attention, concentration, mémoire de travail, langage et orientation dans le temps et l'espace. Les épreuves qui y sont proposées sont souvent plus complexes que celles retrouvées dans le MMSE. Dans le contexte de l'évaluation plus globale de la personne âgée, les qualités métrologiques essentielles



pour la fonction de dépistage de l'outil sont la sensibilité et la spécificité. L'évaluateur voudra s'assurer de dépister toutes les personnes atteintes, sans faux positifs. La cotation de l'évaluation se fait directement sur la grille et simultanément à la passation. L'évaluateur doit inscrire les réponses de la personne et les coter, bon pour un point et incorrect pour 0 point. Un score maximal sur 30 points sera ainsi obtenu. Le score seuil proposé pour distinguer les personnes atteintes des personnes n'ayant pas d'atteinte neurocognitive est de 26/30.

#### 15.7 STROOP

Le Stroop Victoria est une des nombreuses tâches d'évaluation de l'inhibition basée sur l'effet d'interférence proposé par J.R. Stroop (1935) ; ce matériel a pour objectif de fournir aux cliniciens un outil d'évaluation des processus d'inhibition.

La version originale du Stroop Victoria a été proposée en 1991 (Spreen & Strauss, 1991). Une ligne d'exemple pour chaque planche a été ajoutée afin de s'assurer d'une bonne compréhension des consignes par le sujet avant l'administration de la tâche.

Le matériel de l'épreuve se compose de trois planches correspondant à trois conditions, chacune comportant une ligne de dix exemples et dix lignes de stimuli de couleur ou non.

La planche 1 (DENOMINATION [de couleur]) est constituée de petites barres de couleur arrangées en lignes que le sujet doit dénommer. Couleurs : Vert, Bleu, Rouge.

La planche 2 (LECTURE) se compose de mots sans couleur, correspondant aux trois couleurs préalablement présentées : « VERT », « BLEU », « ROUGE ». La tâche du sujet est de lire tout simplement les mots écrits.

Pour la planche 3 (INTERFERENCE), le nom des trois couleurs est écrit avec une encre de couleur différente (par exemple : vert est écrit en rouge). La tâche du sujet est de nommer la couleur de l'encre de chaque mot (et non lire le mot écrit).

Durée totale de passation : 20 minutes.

Hétéroévaluation



| Dénomination | |
|--------------|---------------------------------------------------------|
| Lecture | ROUGE BLEU ROUGE VERT BLEU ROUGE VERT BLEU ROUGE BLEU |
| | ROUGE VERT BLEU ROUGE VERT ROUGE BLEU VERT BLEU VERT |
| | ROUGE BLEU ROUGE VERT BLEU ROUGE VERT BLEU ROUGE BLEU |
| | BLEU VERT ROUGE BOUGE BLEU VERT ROUGE BLEU ROUGE VERT |
| | VERT ROUGE BLEU. VERT ROUGE BLEU HOUGE BLEU. VERT BLEU. |
| | VERT BLEU ROUGE BLEU VERT ROUGE VERT BLEU VERT ROUGE |
| | ROUGE BLEU BLEU ROUGE VERT BLEU VERT BLEU ROUGE VERT |
| | VERT ROUGE VERT BLEU ROUGE VERT ROUGE BLEU VERT ROUGE |
| | ROUGE VERT BLEU ROUGE VERT ROUGE BLEU VERT BLEU ROUGE |
| | BLEU VERT ROUGE VERT ROUGE BLEU ROUGE VERT BLEU ROUGE |
| Interférence | ROUGE BLEU VERT ROUGE BLED ROUGE VERT VERT BLEU BLEU |
| | HOUGE BLEU VERT BLEU HOUGE VERT HOUGE BLEU YERT HOUGE |
| | ROUGE VEHT BLEW ROUGE VEHT ROUGE BLEW VERT ROUGE VEHT |
| | VERT HOUSE BLEU VERT BLEU VERT HOUSE BLEU BLEU BOUSE |
| | ROUGE VERY BLEU VERY ROUGE VERY BLEU ROUGE BLEU VERY |
| | BLEU VERY BLEU ROUGE BLEU ROUGE VERY BLEU ROUGE VERY |
| | VERT ROUGE BLEU ROUGE VERT BLEU ROUGE POUGE VERT BLEU |
| | BLEV ROUGE BLEW VERT ROUGE BLEW VERT ROUGE BLEW HOUGE |
| | VERT BLEU VERT BLEU HOUGE VERT HOUGE BLEU VERT HOUGE |
| | BLEU ROUGE BLEU VERY ROUGE BLEU VERY ROUGE BLEU ROUGE |